CLINICAL TRIAL: NCT03416179
Title: A RANDOMIZED (1:1), DOUBLE-BLIND, MULTI-CENTER, PLACEBO CONTROLLED STUDY EVALUATING INTENSIVE CHEMOTHERAPY WITH OR WITHOUT GLASDEGIB (PF-04449913) OR AZACITIDINE (AZA) WITH OR WITHOUT GLASDEGIB IN PATIENTS WITH PREVIOUSLY UNTREATED ACUTE MYELOID LEUKEMIA
Brief Title: A Study Evaluating Intensive Chemotherapy With or Without Glasdegib or Azacitidine With or Without Glasdegib In Patients With Previously Untreated Acute Myeloid Leukemia
Acronym: BRIGHT AML1019
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B1371019; 2017-002822-19 (EudraCT Number); BRIGHT (Other: Alias Study Number); BRIGHT AML1019 (Other: Alias Study Number)
Record Dates: First submitted 2017-12-21; First posted 2018-01-31 (Actual); Results first posted 2021-06-25 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: glasdegib;; untreated;; Hedgehog Inhibitor
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — glasdegib; Daunorubicin; Cytarabine; Azacitidine

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, multi-center, placebo controlled study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A (Intensive Study) (Experimental): Glasdegib + '7+3' Induction(s)
  Interventions: Drug: glasdegib; Drug: daunorubicin + cytarabine; Drug: cytarabine; Procedure: HSCT
- Arm B (Intensive Study) (Placebo Comparator): Placebo + '7+3' Induction(s)
  Interventions: Drug: daunorubicin + cytarabine; Drug: Placebo; Drug: cytarabine; Procedure: HSCT
- Arm A (Non-intensive study) (Experimental): Glasdegib + azacitidine
  Interventions: Drug: azacitidine; Drug: glasdegib
- Arm B (Non-intensive study) (Placebo Comparator): Placebo + azacitidine
  Interventions: Drug: azacitidine; Drug: Placebo

INTERVENTIONS:
Drug: glasdegib — Daily Glasdegib (100 mg, PO), beginning on Day 1 and is to continue up to 2 years post randomization.
  Following consolidation therapy, glasdegib or placebo will be administered daily for up to 2 years after randomization or until they have minimal residual disease (MRD) negative disease, whichever comes first.
  Daily Glasdegib (100 mg, PO) or matching placebo will continue throughout Induction(s) and Consolidation therapies regardless of dose modifications/delays in the chemotherapy.
  Other Names: PF-04449913
  Arms: Arm A (Intensive Study)
Drug: daunorubicin + cytarabine — '7+3' (cytarabine 100 mg/m2, IV for 7 days by continuous infusion and daunorubicin 60 mg/m2 for 3 days).
  If a second induction is needed, Investigators may choose either a 5 day cytarabine continuous infusion plus daunorubicin for 2 days ('5+2') or a 7 day cytarabine continuous infusion plus daunorubicin for 3 days ('7+3');
  Arms: Arm A (Intensive Study); Arm B (Intensive Study)
Drug: azacitidine — Azacitidine (75 mg/m2, SC or IV) daily for 7 days, in 28 day cycles for as long as they do not meet the criteria for disease progression, unacceptable toxicity, consent withdrawal, or death.
  Arms: Arm A (Non-intensive study); Arm B (Non-intensive study)
Drug: Placebo — Matching placebo (PO) given on Day 1 and is to continue up to 2 years post randomization. Following consolidation therapy, placebo will be administered daily for up to 2 years after randomization or until they have MRD negative disease, whichever comes first.
  Daily placebo will continue throughout Induction(s) and Consolidation therapies regardless of dose modifications/delays in the chemotherapy.
  Arms: Arm B (Intensive Study)
Drug: Placebo — Matching placebo (PO) is to be administered by mouth daily beginning on Day 1 of chemotherapy and will continue if subjects demonstrate reasonable evidence of clinical benefit and do not meet the criteria for progression regardless of any delays/modifications in the chemotherapy treatment. Subjects will continue placebo until disease progression, unacceptable toxicity, consent withdrawal, or death, whichever comes first.
  Arms: Arm B (Non-intensive study)
Drug: glasdegib — Glasdegib 100 mg PO QD is to be administered by mouth daily beginning on Day 1 of chemotherapy and will continue if subjects demonstrate reasonable evidence of clinical benefit and do not meet the criteria for progression regardless of any delays/modifications in the chemotherapy treatment.
  Subjects will continue glasdegib until disease progression, unacceptable toxicity, consent withdrawal, or death, whichever comes first.
  Arms: Arm A (Non-intensive study)
Drug: cytarabine — Consolidation with single agent cytarabine 3 g/m2 IV for adults <60 years and 1 g/m2 for adults 60 years over 3 BID on Days 1, 3, and 5, every 28 days for up to 4 cycles or alternative single agent cytarabine consolidation schedules may be used per local prescribing information.
  Arms: Arm A (Intensive Study); Arm B (Intensive Study)
Procedure: HSCT — If required, and done per standard of care post Induction(s).
  Arms: Arm A (Intensive Study); Arm B (Intensive Study)

SUMMARY:
Glasdegib is being studied in combination with azacitidine for the treatment of adult patients with previously untreated acute myeloid leukemia (AML) who are not candidates for intensive induction chemotherapy (Non-intensive AML population).

Glasdegib is being studied in combination with cytarabine and daunorubicin for the treatment of adult patients with previously untreated acute myeloid leukemia (Intensive AML population).

DETAILED DESCRIPTION:
Two separate registration trials conducted under one protocol number are proposed to adequately and independently evaluate the addition of glasdegib in intensive and non-intensive chemotherapy populations. Each study will have an experimental treatment arm and a placebo arm. Endpoints are the same for each study except where specifically indicated.

Assignment to the Intensive Study or the Non-Intensive Study will be made by the Investigator based on the 2017 European LeukemiaNet (ELN) recommendations.

Study B1371019 is a randomized (1:1), double-blind, multi-center, placebo controlled study of chemotherapy in combination with glasdegib versus chemotherapy in combination with placebo in adult patients with previously untreated AML.

Glasdegib is being studied in combination with azacitidine for the treatment of adult patients with previously untreated acute myeloid leukemia (AML) who are not candidates for intensive induction chemotherapy (Non-intensive AML population).

Glasdegib is being studied in combination with cytarabine and daunorubicin for the treatment of adult patients with previously untreated acute myeloid leukemia (Intensive AML population).

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the Intensive and Non Intensive study (unless where indicated):

1. Subjects with untreated AML according to the World Health Organization (WHO) 2016 Classification2, including those with:

   * AML arising from MDS or another antecedent hematologic disease (AHD).
   * AML after previous cytotoxic therapy or radiation (secondary AML).
2. 18 years of age (In Japan, 20 years of age).
3. Adequate Organ Function as defined by the following:

   * Serum aspartate aminotransferase (AST) and serum alanine aminotransferase (ALT) 3 x upper limit of normal (ULN), excluding subjects with liver function abnormalities due to underlying malignancy.
   * Total serum bilirubin 2 x ULN (except subjects with documented Gilbert's syndrome).
   * Estimated creatinine clearance 30 mL/min as calculated using the standard method for the institution.
4. QTc interval 470 msec using the Fridericia correction (QTcF).
5. All anti cancer treatments (unless specified) should be discontinued 2 weeks from study entry, for example: targeted chemotherapy, radiotherapy, investigational agents, hormones, anagrelide or cytokines.

   * For control of rapidly progressing leukemia, all trans retinoic acid (ATRA), hydroxyurea, and/or leukopheresis may be used before and for up to 1 week after the first dose of glasdegib.
6. Serum or urine pregnancy test (for female subjects of childbearing potential) with a minimum sensitivity of 25 IU/L or equivalent units of human chorionic gonadotropin (hCG) negative at screening.
7. Male and female subjects of childbearing potential and at risk for pregnancy must agree to use at least one highly effective method of contraception throughout the study and for 180 days after the last dose of azacitidine, cytarabine, or daunorubicin; and the last dose of glasdegib or placebo, whichever occurs later.
8. Female subjects of non childbearing potential must meet at least 1 of the following criteria:

   1. Have undergone a documented hysterectomy and/or bilateral oophorectomy;
   2. Have medically confirmed ovarian failure; or
   3. Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; status may be confirmed by having a serum follicle stimulating hormone (FSH) level confirming the postmenopausal state.

   All other female subjects (including female subjects with tubal ligations) are considered to be of childbearing potential.
9. Consent to a saliva sample collection for a germline comparator, unless prohibited by local regulations or ethics committee (EC) decision.
10. Evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study.
11. Subjects who are willing and able to comply with the study scheduled visits, treatment plans, laboratory tests and other procedures (including bone marrow [BM] assessments).

Exclusion Criteria:

Subjects with any of the following characteristics/conditions will not be included in the study:

1. Acute Promyelocytic Leukemia (APL) and APLwith PML RARA, subjects (WHO 2016 classification).
2. AML with BCR ABL1 or t(9;22)(q34;q11.2) as a sole abnormality.

   * Complex genetics may include t(9;22) cytogenetic translocation.
3. Subjects with known active CNS leukemia.
4. Participation in other clinical studies involving other investigational drug(s) (Phases 1 4) within 4 weeks prior study entry and/or during study participation.
5. Subjects known to be refractory to platelet or packed red cell transfusions per Institutional Guidelines, or a patient who refuses blood product support.
6. Subjects with another active malignancy on treatment with the exception of basal cell carcinoma, non melanoma skin cancer, cervical carcinoma in situ. Other prior or concurrent malignancies will be considered on a case by case basis.
7. Any one of the following ongoing or in the previous 6 months: myocardial infarction, congenital long QT syndrome, Torsades de pointes, symptomatic arrhythmias (including sustained ventricular tachyarrhythmia), right or left bundle branch block and bifascicular block, unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure (CHF New York Heart Association class III or IV), cerebrovascular accident, transient ischemic attack or symptomatic pulmonary embolism; as well as bradycardia defined as <50 bpms.
8. Subjects with an active, life threatening or clinically significant uncontrolled systemic infection not related to AML.
9. Subjects with left ventricular ejection fraction (LVEF) <50% are excluded from the Intensive Chemotherapy Study only.
10. Cumulative anthracycline dose equivalent of 550 mg/m2 of daunorubicin for the Intensive Chemotherapy Study only.
11. Known malabsorption syndrome or other condition that may significantly impair absorption of study medication in the investigator's judgment (eg, gastrectomy, lap band, Crohn's disease) and inability or unwillingness to swallow tablets or capsules.
12. Current use or anticipated requirement for drugs that are known strong CYP3A4/5 inducers.
13. Concurrent administration of herbal preparations.
14. Major surgery or radiation within 4 weeks of starting study treatment.
15. Documented or suspected hypersensitivity to any one of the following:

    * For subjects assigned to intensive chemotherapy, documented or suspected hypersensitivity to cytarabine (not including drug fever or exanthema, including known cerebellar side effects) or daunorubicin.
    * For subjects assigned to non intensive chemotherapy, documented or suspected hypersensitivity to azacitidine or mannitol.
16. Known active drug or alcohol abuse.
17. Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
18. Pregnant females or breastfeeding female subjects.
19. Known recent or active suicidal ideation or behavior.
20. Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or subjects who are Pfizer employees, including their family members, directly involved in the conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 730 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2022-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (149):
- United States (30):
  - UCLA Department of Medicine, Los Angeles, California
  - UCLA Drug Information/Investigational Drugs, Los Angeles, California
  - UCLA Hematology/Oncology Clinic, Los Angeles, California
  - UCLA Ronald Reagan Medical Center, Los Angeles, California
  - UC Irvine Health - Chao Family Comprehensive Cancer Center, Orange, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - University of California, San Francisco, San Francisco, California
  - UCLA Hematology/Oncology - Westlake Village, Westlake Village, California
  - Augusta University Medical Center, Augusta, Georgia
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - Tufts Medical Center Investigational Drug Pharmacy, Boston, Massachusetts
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - MidAmerica Division, Inc., c/o Research Medical Center, Kansas City, Missouri
  - Northwell Health/Monter Cancer Center, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - University of Rochester Medical Center, Rochester, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - OHSU Center for Health and Healing, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Centennial Medical Center, Nashville, Tennessee
  - TriStar Bone Marrow Transplant, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - Blood Cancer and Stem Cell Transplant Clinic, San Antonio, Texas
  - Methodist Healthcare System of San Antonio, San Antonio, Texas
  - Swedish Cancer Institute, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
- Australia (3):
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
- Austria (3):
  - Landeskrankenhaus Salzburg, Universitatsklinik fur Innere Medizin III der PMU, Salzburg
  - Uniklinikum Salzburg, Landeskrankenhaus Salzburg, Salzburg
  - Krankenhaus Hietzing mit Neurologischem Zentrum Rosenhugel, Vienna
- Belgium (4):
  - AZ Sint-Jan Brugge-Oostende av, Bruges
  - Universitaire Ziekenhuizen Brussel (UZ Brussel), Brussels
  - Universitaire Ziekenhuizen Brussel, Brussels
  - Universitaire Ziekenhuizen Leuven, Leuven
- Canada (7):
  - Health Sciences Centre, Winnipeg, Manitoba
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Sunnybrook Research Institute, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - CIUSSS de l'Est-de-l'Ile-de- Montréal - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- China (13):
  - The First Affiliated Hospital of USTC, Anhui Provincial Hospital, Hefei, Anhui
  - Anhui Provincial Hospital, Hefei, Anhui
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Guangdong Second Provincial General Hospital, Guangzhou, Guangdong
  - Hebei Yanda Lu Daopei Hospital, Langfang, Hebei
  - Henan Provincial People's Hospital/Hematology Department, Zhengzhou, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology/Cancer Center, Wuhan, Hubei
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital College of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Ruijin Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai
- Czechia (6):
  - Interni hematologicka a onkologicka klinika, Fakultni nemocnice Brno, Brno
  - Nemocnicni lekarna, Brno
  - Ustavni lekarna, Ostrava - Poruba
  - Klinika hematoonkologie, Ostrava-Poruba
  - Interní hematologická klinika, Fakultni nemocnice Královské Vinohrady, Prague
  - Ústavni lékárna, Prague
- France (6):
  - CHU Henri Mondor, Créteil
  - CHU de Nantes Hotel Dieu, Nantes
  - CHU de Nantes, Nantes
  - Hopital Saint Louis, Paris
  - Centre Hospitalier Lyon Sud - Service d'Hematologie, Pierre-Bénite
  - Institut Gustave Roussy, Villejuif
- Germany (6):
  - Klinikum der Universitaet Muenchen, Munich, Bavaria
  - Philipps-Universitaet Marburg, Marburg, Hesse
  - Universitätsklinikum Köln, Cologne, North Rhine-Westphalia
  - Universitaetsklinikum Muenster, Münster, North Rhine-Westphalia
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
- Hungary (6):
  - Debreceni Egyetem Klinikai Kozpont Belgyogyaszati Klinika, Hematologia Tanszek, Debrecen
  - Debreceni Egyetem Klinikai Kozpont Belgyogyaszati Klinika, Debrecen
  - Petz Aladár Megyei Oktató Kórház, II. Belgyógyászat- Hematológiai Osztály, Győr
  - Somogy Megyei Kaposi Mor Oktato Korhaz, Kaposvár
  - Szabolcs-Szatmar Bereg Megyei Korhazak es Egyetemi Oktatokorhaz, Josa Andras Korhaz, Hematologia, Nyíregyháza
  - Szabolcs-Szatmar Bereg Megyei Korhazak es Egyetemi Oktatokorhaz, Josa Andras Korhaz,, Nyíregyháza
- Israel (5):
  - Rambam Health Care Campus, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Medical Center (Ein Kerem), Jerusalem
  - Hemato-oncology ambulatory Service, Petah Tikva
  - Rabin Medical Center, Beilinson Hospital, Petah Tikva
- Italy (7):
  - AOU Ospedali Riuniti Umberto I, G.M. Lancisi, G. Salesi, Clinica Di Ematologia, Torrette Di Ancona, Ancona
  - SOD Farmacia-Dipt dei servizi -AOU Ospedali Riuniti Umberto I, G.M. Lancisi, G. Salesi, Torette Di Ancona, AN
  - A.O.U. di Ferrara- Arcispedale Sant'Anna,, Cona, Ferrara, FE
  - AO Ospedali Riuniti Marche Nord - Presidio Ospedaliero San Salvatore di Pesaro -, Pesaro, PU
  - Azienda Ospedaliera Universitaria Senese., Siena, SI
  - Azienda Ospedaliero Universitaria di Bologna Policlinico S.Orsola Malpighi, Bologna
  - Azienda Ospedaliera Universitaria Senese, Siena
- Japan (15):
  - Japanese Red Cross Nagoya Daini Hospital, Nagoya, Aichi-ken
  - University of Fukui Hospital, Yoshida-gun, Fukui
  - Gunma University Hospital, Maebashi, Gunma
  - Kobe University Hospital, Kobe, Hyōgo
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Tohoku University Hospital, Sendai, Miyagi
  - Osaka City University Hospital, Osaka, Osaka
  - Kindai University Hospital, Ōsaka-sayama, Osaka
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - National Hospital Organization Disaster Medical Center, Tachikawa, Tokyo
  - Akita University Hospital, Akita
  - Kyushu University Hospital, Fukuoka
  - National Hospital Organization Kumamoto Medical Center, Kumamoto
  - Nagasaki University Hospital, Nagasaki
  - Tokyo Medical University Hospital, Tokyo
- Mexico (2):
  - Instituto Nacional de Cancerología, México, MÉX
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey, Nuevo León
- Poland (2):
  - Klinika Hematologii i Transplantologii Uniwersyteckie Centrum Kliniczne, Gdansk
  - WWCOiT im. M. Kopernika w Lodzi, Lodz
- Romania (4):
  - Institutul Oncologic 'Prof. Dr. Ion Chiricuta', Cluj-Napoca, Cluj
  - Spitalul Clinic Municipal Filantropia Craiova, Sectia Clinica Hematologie, Craiova, Dolj
  - Sp. Clinic de Urgenta Militar Central Dr. Carol Davila, Bucharest
  - Spitalul Clinic Coltea, Clinica de Hematologie, Bucharest
- Russia (4):
  - State Budgetary Healthcare Institution of Moscow, Moscow
  - SBHI NNR NN RCH n. a. N.A. Semashko, Nizhny Novgorod
  - State Budgetary Institution of Ryazan Region 'Regional Clinical Hospital' (SBI RR RCH), Ryazan
  - V.A Almazov NMRC, Saint Petersburg
- South Korea (9):
  - Chonbuk National University Hospital, Jeonju, Jeollabuk-do
  - Inje University Busan Paik Hospital, Busan
  - Keimyung University Dongsan Hospital, Daegu
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Hospital, Seoul
  - Clinical Trial Center, Severance Hospital, Yonsei University Health System, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul
- Spain (7):
  - Hospital del Mar, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Arnau de Vilanova, Lleida
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
- Sweden (2):
  - Universitetssjukhuset Orebro, Örebro
  - Karolinska Universitetssjukhuset Huddinge, Stockholm
- Taiwan (5):
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - Chang Gung Memorial Hospital-Linkou Branch, Taoyuan
- United Kingdom (3):
  - The Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham, WEST Midlands
  - Imperial College Healthcare NHS Trust, London

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Sekeres MA, Montesinos P, Novak J, Wang J, Jeyakumar D, Tomlinson B, Mayer J, Jou E, Robak T, Taussig DC, Dombret H, Merchant A, Shaik N, O'Brien T, Roh W, Liu X, Ma W, DiRienzo CG, Chan G, Cortes JE. Glasdegib plus intensive or non-intensive chemotherapy for untreated acute myeloid leukemia: results from the randomized, phase 3 BRIGHT AML 1019 trial. Leukemia. 2023 Oct;37(10):2017-2026. doi: 10.1038/s41375-023-02001-z. Epub 2023 Aug 21. PMID 37604981
- [Derived] Cortes JE, Dombret H, Merchant A, Tauchi T, DiRienzo CG, Sleight B, Zhang X, Leip EP, Shaik N, Bell T, Chan G, Sekeres MA. Glasdegib plus intensive/nonintensive chemotherapy in untreated acute myeloid leukemia: BRIGHT AML 1019 Phase III trials. Future Oncol. 2019 Nov;15(31):3531-3545. doi: 10.2217/fon-2019-0373. Epub 2019 Sep 13. PMID 31516032
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B1371019

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study evaluated glasdegib in intensive and non-intensive chemotherapy populations. Intensive study: Glasdegib was studied in combination with cytarabine and daunorubicin for the treatment of adult participants with previously untreated acute myeloid leukemia (AML). Non-intensive study: Glasdegib was studied in combination with azacitidine for the treatment of adult participants with previously untreated AML who were not candidates for intensive induction chemotherapy.
Pre-assignment Details: Inadvertently 1 participant was enrolled twice into the study resulting in enrollment number as 730. However, a total of 729 participants were randomized and received treatment in the study.
  Although participation of participants was terminated by the sponsor, the study was considered completed as participants were fully enrolled as planned.
Groups:
- Intensive Study: Glasdegib + Cytarabine + Daunorubicin: Participants received first induction therapy (28 days) (backbone chemotherapy+experimental therapy). Backbone chemotherapy: Cytarabine 100 milligram per square meter (mg/m^2) daily by intravenous (IV) infusion for 7 days along with daunorubicin 60 mg/m^2 daily IV for 3 days. Depending upon bone marrow blast or investigator judgement participants had second induction i.e. received either same backbone therapy or cytarabine 100 mg/m^2 IV daily for 5 days and daunorubicin 60 mg/m^2 IV daily for 2 days. Participants with less than (<) 5% bone marrow blasts entered into consolation phase- treated with either or both of following: 1) cytarabine 1 to 3 gram per square meter (gm/m^2) IV for adults greater than or equals to (>=) 60 to <60 years twice daily on Days 1, 3, and 5 for 4 cycle (each cycle 28 day) or cytarabine per local prescribing information. 2) Received hematopoietic stem cell transplantation (HSCT) per local standard of care. Experimental Therapy: Participants were to receive Glasdegib 100 milligram (mg) tablet orally (PO) once daily (QD) from Day 1 of chemotherapy up to 28 days in both induction until 2 consecutive complete remission (CR) minimal residual disease (MRD)-negative central laboratory results, whichever came first (1.6 year).
- Intensive Study: Placebo + Cytarabine + Daunorubicin: Participants received first induction therapy (28 days) (backbone chemotherapy+experimental therapy). Backbone chemotherapy: Cytarabine 100 mg/m^2 daily by IV infusion for 7 days along with daunorubicin 60 mg/m^2 daily IV for 3 days. Depending upon bone marrow blast or investigator judgement participants had second induction i.e. received either same backbone therapy or cytarabine 100 mg/m^2 IV daily for 5 days and daunorubicin 60 mg/m^2 IV daily for 2 days. Participants with <5% bone marrow blasts entered into consolation phase- treated with either or both of following: 1) cytarabine 1 to 3 gram/m^2 IV for adults >=60 to <60 years twice daily on Days 1, 3, and 5 for 4 cycle (each cycle 28 day) or cytarabine per local prescribing information. 2) Received HSCT per local standard of care. Experimental Therapy: Participants were to receive Glasdegib 100 mg matching placebo tablet PO QD from Day 1 of chemotherapy up to 28 days in both induction until 2 consecutive CR MRD-negative central laboratory results, whichever came first (1.8 year).
- Non-intensive Study: Glasdegib + Azacitidine: Participants received chemotherapy with azacitidine 75 mg/m^2 SC injection or IV infusion from Day 1 up to Day 7 of each cycle (28 day) and continued for at least 6 cycles or until unacceptable toxicity, participant refusal or death, whichever occurred first. Participants also were to receive glasdegib 100 mg PO QD from Day 1 of chemotherapy until clinical benefit or disease progression, unacceptable toxicity, consent withdrawal, or death, whichever occurred first. Eligible participants underwent HSCT per local standard of care and were to receive glasdegib unless 2 consecutive negative MRD assessments (3 year).
- Non-intensive Study: Placebo + Azacitidine: Participants received chemotherapy with azacitidine 75 mg/m^2 SC injection or IV infusion from Day 1 up to Day 7 of each cycle (28 day) and continued for at least 6 cycles or until unacceptable toxicity, participants refusal or death, whichever occurred first. Participants also received glasdegib 100 mg tablet matching placebo PO QD from Day 1 of chemotherapy until clinical benefit or disease progression, unacceptable toxicity, consent withdrawal, or death, whichever occurred first. Eligible participants underwent HSCT per local standard of care and were to receive glasdegib matching placebo unless 2 consecutive negative MRD assessments (2.44 year).
Period: Overall Study
Arm/Group | Intensive Study: Glasdegib + Cytarabine + Daunorubicin | Intensive Study: Placebo + Cytarabine + Daunorubicin | Non-intensive Study: Glasdegib + Azacitidine | Non-intensive Study: Placebo + Azacitidine
Started | 201 | 203 | 163 | 162
Treated | 198 | 201 | 162 | 160
Completed | 0 | 1 | 13 | 6
Not Completed | 201 | 202 | 150 | 156
Not completed — Death | 90 | 87 | 117 | 113
Not completed — Withdrawal by Subject | 15 | 20 | 6 | 9
Not completed — Lost to Follow-up | 1 | 1 | 0 | 3
Not completed — Study participation terminated by Sponsor | 93 | 91 | 26 | 31
Not completed — Other | 2 | 3 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis (FA) set included all randomized participants.
Groups:
- Intensive Study: Glasdegib + Cytarabine + Daunorubicin: Participants received first induction therapy (28 days) (backbone chemotherapy+experimental therapy). Backbone chemotherapy: Cytarabine 100 mg/m^2 daily by IV infusion for 7 days along with daunorubicin 60 mg/m^2 daily IV for 3 days. Depending upon bone marrow blast or investigator judgement participants had second induction i.e. received either same backbone therapy or cytarabine 100 mg/m^2 IV daily for 5 days and daunorubicin 60 mg/m^2 IV daily for 2 days. Participants with <5% bone marrow blasts entered into consolation phase- treated with either or both of following: 1) cytarabine 1 to 3 gm/m^2 IV for adults >=60 to <60 years twice daily on Days 1, 3, and 5 for 4 cycle (each cycle 28 day) or cytarabine per local prescribing information. 2) Received HSCT per local standard of care. Experimental Therapy: Participants were to receive Glasdegib 100 mg tablet PO QD from Day 1 of chemotherapy up to 28 days in both induction until 2 consecutive CRMRD-negative central laboratory results, whichever came first (1.6 year).
- Total: Total of all reporting groups
Arm/Group | Intensive Study: Glasdegib + Cytarabine + Daunorubicin | Intensive Study: Placebo + Cytarabine + Daunorubicin | Non-intensive Study: Glasdegib + Azacitidine | Non-intensive Study: Placebo + Azacitidine | Total
Number analyzed (Participants) | 201 | 203 | 163 | 162 | 729
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.55 (12.60) | 55.38 (13.61) | 73.19 (7.17) | 73.14 (6.82) | 63.63 (13.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 97 | 97 | 89 | 354
  Male | 130 | 106 | 66 | 73 | 375
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 12 | 12 | 16 | 59
  Not Hispanic or Latino | 166 | 171 | 140 | 139 | 616
  Unknown or Not Reported | 16 | 20 | 11 | 7 | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 66 | 57 | 51 | 44 | 218
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 3 | 1 | 7 | 14
  White | 110 | 123 | 97 | 99 | 429
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 20 | 20 | 14 | 12 | 66

OUTCOME MEASURES:

1. Primary Outcome: Intensive Study: Overall Survival (OS)
Description: OS is defined as the time from the date of randomization to the date of death due to any cause. Participants last known to be alive were to be censored at the date of last contact.
Time Frame: Baseline up to 25 months
Population: FA set included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Intensive Study: Glasdegib + Cytarabine + Daunorubicin | Intensive Study: Placebo + Cytarabine + Daunorubicin
Number analyzed (Participants) | 201 | 203
months | 17.3 [15.2 to 18.5] | 20.4 [17.6 to NA] — Upper limit of 95 % CI was not estimable due to low number of participants with events.
Statistical Analysis 1: Comparison: Intensive Study: Glasdegib + Cytarabine + Daunorubicin vs Intensive Study: Placebo + Cytarabine + Daunorubicin; Hazard ratio based on Cox proportional hazards model; under proportional hazards, hazard ratio less than (<) 1 indicated a reduction in hazard rate in favor of Glasdegib 100 mg PO + Cytarabine 100 mg/m^2 IV + Daunorubicin 60 mg/m^2 compared to Placebo + Cytarabine 100 mg/m^2 IV + Daunorubicin 60 mg/m^2; Test type: Superiority; p = 0.6579, Log Rank; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.755 to 1.532]

2. Primary Outcome: Non-intensive Study: Overall Survival (OS)
Description: as for outcome 1
Time Frame: Baseline up to 25 months
Population: FA set included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Non-intensive Study: Glasdegib + Azacitidine | Non-intensive Study: Placebo + Azacitidine
Number analyzed (Participants) | 163 | 162
months | 10.3 [7.7 to 12.4] | 10.6 [8.4 to 13.3]
Statistical Analysis 1: Comparison: Non-intensive Study: Glasdegib + Azacitidine vs Non-intensive Study: Placebo + Azacitidine; Hazard ratio based on Cox proportional hazards model; under proportional hazards, hazard ratio < 1 indicated a reduction in hazard rate in favor of Glasdegib 100 mg PO QD + Azacitidine compared to Placebo + Azacitidine; Test type: Superiority; p = 0.5955, Log Rank; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.775 to 1.388]

3. Secondary Outcome: Intensive Study: Percentage of Participants Who Improved in Fatigue Score Measured by the MD Anderson Symptom Inventory -Acute Myelogenous Leukemia/Myelodysplastic Syndrome (MDASI-AML/MDS) Questionnaire
Description: MDASI-AML/MDS: consists of 23 items, 13-item core cancer symptoms (pain, fatigue, nausea, disturbed sleep, distress, shortness of breath, problem remembering, lack of appetite, drowsiness, dry mouth, sadness, vomiting, and numbness), 4-item AML/MDS specific symptoms (malaise, diarrhea, muscle weakness, and skin problems), and 6 areas of interference (general activity, mood, work, walking, relations with other people, and enjoyment of life). "Fatigue" was measured at the participants' worst level in last 24 hours by asking participants to respond to each item on an 0-10 numeric rating scale (NRS), where 0 = "not present" and 10 = "as bad as you can imagine". Percentage of participants who had improvement in "fatigue" symptoms reported in this outcome measure.
Time Frame: Post-baseline up to Week 8
Population: FA set included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Intensive Study: Glasdegib + Cytarabine + Daunorubicin | Intensive Study: Placebo + Cytarabine + Daunorubicin
Number analyzed (Participants) | 201 | 203
Percentage of participants | 17.41 [12.17 to 22.66] | 17.24 [12.05 to 22.44]
Statistical Analysis 1: Comparison: Intensive Study: Glasdegib + Cytarabine + Daunorubicin vs Intensive Study: Placebo + Cytarabine + Daunorubicin; Test type: Other; p = 0.5095, Mantel Haenszel

4. Secondary Outcome: Non-intensive Study: Percentage of Participants Who Improved in Fatigue Score Measured by the MDASI-AML/MDS Questionnaire at Week 12
Description: MDASI-AML/MDS: consists of 23 items, 13-item core cancer symptoms (pain, fatigue, nausea, disturbed sleep, distress, shortness of breath, problem remembering, lack of appetite, drowsiness, dry mouth, sadness, vomiting, and numbness), 4-item AML/MDS specific symptoms (malaise, diarrhea, muscle weakness, and skin problems), and 6 areas of interference (general activity, mood, work, walking, relations with other people, and enjoyment of life). "Fatigue" was measured at the participants' worst level in last 24 hours by asking participants to respond to each item on an 0-10 NRS, where 0 = "not present" and 10 = "as bad as you can imagine". Percentage of participants who had improvement in "fatigue" symptoms reported in this outcome measure.
Time Frame: Post-baseline up to Week 12
Population: FA set included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Non-intensive Study: Glasdegib + Azacitidine | Non-intensive Study: Placebo + Azacitidine
Number analyzed (Participants) | 163 | 162
Percentage of participants | 11.66 [6.73 to 16.58] | 15.43 [9.87 to 21.00]
Statistical Analysis 1: Comparison: Non-intensive Study: Glasdegib + Azacitidine vs Non-intensive Study: Placebo + Azacitidine; Test type: Other; p = 0.8359, Mantel Haenszel

5. Secondary Outcome: Intensive Study: Percentage of Participants With Complete Remission Without Negative Minimal Residual Disease (CRMRD-neg)
Description: Complete remission (CR) was defined based on 2017 European LeukemiaNet (ELN) recommendations. CR: Bone marrow blasts <5 percentage (%); absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count (ANC) greater than equal to (>=) 1.0*10^9/Liter (L); platelet count >=100*10^9/L. CRMRD-neg: CR with negativity for a genetic marker by reverse transcription quantitative polymerase chain reaction (RT-qPCR), or CR with negativity by Multiparameter Flow Cytometry (MFC).
Time Frame: Day 1 up to maximum of 2 years
Population: FA set included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Intensive Study: Glasdegib + Cytarabine + Daunorubicin | Intensive Study: Placebo + Cytarabine + Daunorubicin
Number analyzed (Participants) | 201 | 203
Percentage of participants | 5.0 [2.4 to 9.0] | 5.4 [2.7 to 9.5]

6. Secondary Outcome: Non-intensive Study: Percentage of Participants With Complete Remission Without Negative Minimal Residual Disease (CRMRD-neg)
Description: CR was defined based on 2017 ELN recommendations. CR: Bone marrow blasts <5%; absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease; ANC >=1.0*10^9/L; platelet count >=100*10^9/L. CRMRDneg: CR with negativity for a genetic marker by RT-qPCR, or CR with negativity by MFC.
Time Frame: Day 1 up to maximum of 3 years
Population: FA set included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Non-intensive Study: Glasdegib + Azacitidine | Non-intensive Study: Placebo + Azacitidine
Number analyzed (Participants) | 163 | 162
Percentage of participants | 1.8 [0.4 to 5.3] | 0.6 [0.0 to 3.4]

7. Secondary Outcome: Intensive Study: Percentage of Participants With Complete Remission Including Negative Minimal Residual Disease (CRMRD-neg)
Description: as for outcome 6
Time Frame: Day 1 up to maximum of 2 years
Population: FA set included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Intensive Study: Glasdegib + Cytarabine + Daunorubicin | Intensive Study: Placebo + Cytarabine + Daunorubicin
Number analyzed (Participants) | 201 | 203
Percentage of participants | 49.3 [42.1 to 56.4] | 47.3 [40.3 to 54.4]

8. Secondary Outcome: Non-intensive Study: Percentage of Participants With Complete Remission (CR) Including Negative Minimal Residual Disease (CRMRD-neg)
Description: as for outcome 6
Time Frame: Day 1 up to maximum of 3 years
Population: FA set included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Non-intensive Study: Glasdegib + Azacitidine | Non-intensive Study: Placebo + Azacitidine
Number analyzed (Participants) | 163 | 162
Percentage of participants | 19.6 [13.8 to 26.6] | 13.0 [8.2 to 19.1]

9. Secondary Outcome: Intensive Study: Percentage of Participants With Complete Remission With Incomplete Hematologic Recovery (CRi)
Description: CR was defined based on 2017 ELN recommendations. CR: MRD (positive or unknown), bone marrow blasts <5%; absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease; ANC less than (<) 1.0*10^9/L; platelet count <100 × 10^9/L. CRi (included CR [includes CRMRD-neg]): not qualifying for CR, neutropenia <1.0*10^9/L or platelets <100*10^9, absence of extramedullary disease, and absence of blasts with Auer rods.
Time Frame: Day 1 up to maximum of 2 years
Population: FA set included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Intensive Study: Glasdegib + Cytarabine + Daunorubicin | Intensive Study: Placebo + Cytarabine + Daunorubicin
Number analyzed (Participants) | 201 | 203
Percentage of participants | 1.5 [0.3 to 4.3] | 5.4 [2.7 to 9.5]

10. Secondary Outcome: Non-intensive Study: Percentage of Participants With Complete Remission With Incomplete Hematologic Recovery (CRi)
Description: CR was defined based on 2017 ELN recommendations. CR: MRD (positive or unknown), bone marrow blasts <5%; absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease; ANC <1.0*10^9/L; platelet count <100 × 10^9/L. CRi (included CR [includes CRMRD-neg]): not qualifying for CR, neutrophil <0.5*10^9/L or platelets <50*10^9, absence of extramedullary disease, and absence of blasts with Auer rods.
Time Frame: Day 1 up to maximum of 3 years
Population: FA set included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Non-intensive Study: Glasdegib + Azacitidine | Non-intensive Study: Placebo + Azacitidine
Number analyzed (Participants) | 163 | 162
Percentage of participants | 2.5 [0.7 to 6.2] | 4.9 [2.2 to 9.5]

11. Secondary Outcome: Intensive Study: Percentage of Participants With Morphologic Leukemia-free State (MLFS)
Description: MLFS was defined based on 2017 ELN recommendations. MLFS: MRD (positive or unknown), bone marrow blasts <5%, no hematologic recovery required, marrow should not be aplastic, at least 200 cells enumerated or cellularity absence of extramedullary disease >=10%, and absence of blasts with Auer rods.
Time Frame: Day 1 up to maximum of 2 years
Population: FA set included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Intensive Study: Glasdegib + Cytarabine + Daunorubicin | Intensive Study: Placebo + Cytarabine + Daunorubicin
Number analyzed (Participants) | 201 | 203
Percentage of participants | 1.5 [0.3 to 4.3] | 2.0 [0.5 to 5.0]

12. Secondary Outcome: Non-intensive Study: Percentage of Participants With Morphologic Leukemia-free State (MLFS)
Description: as for outcome 11
Time Frame: Day 1 up to maximum of 3 years
Population: FA set included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Non-intensive Study: Glasdegib + Azacitidine | Non-intensive Study: Placebo + Azacitidine
Number analyzed (Participants) | 163 | 162
Percentage of participants | 3.1 [1.0 to 7.0] | 0.6 [0.0 to 3.4]

13. Secondary Outcome: Intensive Study: Percentage of Participants With Partial Remission (PR)
Description: PR was defined based on 2017 ELN recommendations. PR: MRD (positive or unknown); bone marrow blasts - decrease to 5-25% and decrease of pre-treatment bone marrow blast percentage by at least 50%; neutrophil count >=1.0*10^9/L; and platelets count >=100*10^9/L.
Time Frame: Day 1 up to maximum of 2 years
Population: FA set included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Intensive Study: Glasdegib + Cytarabine + Daunorubicin | Intensive Study: Placebo + Cytarabine + Daunorubicin
Number analyzed (Participants) | 201 | 203
Percentage of participants | 5.0 [2.4 to 9.0] | 4.4 [2.0 to 8.2]

14. Secondary Outcome: Non-intensive Study: Percentage of Participants With Partial Remission (PR)
Description: as for outcome 13
Time Frame: Day 1 up to maximum of 3 years
Population: FA set included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Non-intensive Study: Glasdegib + Azacitidine | Non-intensive Study: Placebo + Azacitidine
Number analyzed (Participants) | 163 | 162
Percentage of participants | 2.5 [0.7 to 6.2] | 4.9 [2.2 to 9.5]

15. Secondary Outcome: Non-intensive Study: Percentage of Participants With Complete Remission With Partial Hematologic Recovery (CRh)
Description: CRh: MRD (positive or unknown); bone marrow blasts <5%; assessed in non-intensive chemotherapy study only, not qualifying for CR, ie, both neutrophil >=0.5*10^9/L and platelets >=50*10^9/L must be met, but does not satisfy both neutrophils >=1*10^9/L and platelets >=100*10^9/L at the same time; absence of extramedullary disease; and absence of blasts with Auer rods.
Time Frame: Day 1 up to maximum of 3 years
Population: FA set included all randomized participants. This outcome measure was planned to be analyzed only in non-intensive study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Non-intensive Study: Glasdegib + Azacitidine | Non-intensive Study: Placebo + Azacitidine
Number analyzed (Participants) | 163 | 162
Percentage of participants | 3.1 [1.0 to 7.0] | 3.1 [1.0 to 7.1]

16. Secondary Outcome: Intensive Study: Duration of Response (DoRi)
Description: DoRi: only defined for participants who have ever achieved CRi or better (included CR as well) on study as the time from date of first achieving CRi or better to the date of relapse after CRi or better or death due to any cause. CRi: not qualifying for CR, neutropenia <1.0*10^9/L or platelets <100*10^9, absence of extramedullary disease, and absence of blasts with Auer rods. CR was defined based on 2017 ELN recommendations. CR: Bone marrow blasts <5 %; absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease; ANC >=1.0*10^9/L; platelet count >=100*10^9/L. Participants last known to be alive who were free from relapse after CRi or better were censored at the date of last disease assessment that verifies their status.
Time Frame: From date of first achieving CRi or better to the date of relapse after CRi or better or death due to any cause (maximum up to 2 years)
Population: The intensive cohort was terminated because of futility. Participants ended study intervention early and were not followed up as planned. Hence, DORi was not collected, analyzed and reported.
Arm/Group | Intensive Study: Glasdegib + Cytarabine + Daunorubicin | Intensive Study: Placebo + Cytarabine + Daunorubicin
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Non-intensive Study: Duration of Response (DoRi) or (DoRh)
Description: DoRi: only defined for participants who have ever achieved CRi or better (included CR and CRh) on study as the time from date of first achieving CRi or better to the date of relapse after CRi or better or death due to any cause. DoRh: participants who had ever achieved CRh or better (included CR) on study as the time from date of first achieving CRh or better to the date of disease progression, or relapse after CRh or better, or death due to any cause. CRi: not qualifying for CR, neutrophil <0.5*10^9/L or platelets <50*10^9, absence of extramedullary disease, and absence of blasts with Auer rods. CRh: MRD (positive or unknown); bone marrow blasts <5%; assessed in non-intensive chemotherapy study only, not qualifying for CR, ie, both neutrophil >=0.5*10^9/L and platelets >=50*10^9/L must be met, but does not satisfy both neutrophils >=1*10^9/L and platelets >=100*10^9/L at the same time; absence of extramedullary disease; and absence of blasts with Auer rods.
Time Frame: From date of first achieving CRi/CRh or better to the date of relapse/disease progression after CRi/CRh or better or death due to any cause (maximum up to 3 years)
Population: The non-intensive cohort was terminated because of futility. Participants ended study intervention early and were not followed up as planned. Hence, DORi and DoRh was not collected, analyzed and reported.
Arm/Group | Non-intensive Study: Glasdegib + Azacitidine | Non-intensive Study: Placebo + Azacitidine
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Non-intensive Study: Time to Response
Description: TTRi:Participants who achieved CRi or better, as the time from date of randomization to first documentation of response(CRi or better).TTRh:Participants who achieved CRh or better, as the time from date of randomization to first documentation of response(CRh or better). CRi:not qualifying for CR, neutrophil<0.5*10^9/L or platelets<50*10^9, absence of extramedullary disease,absence of blasts with Auer rods. CR was defined based on 2017 ELN recommendations. CR: Bone marrow blasts <5 %; absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease; ANC >=1.0*10^9/L; platelet count >=100*10^9/L. CRh: MRD (positive or unknown); bone marrow blasts <5%; assessed in non-intensive chemotherapy study only, not qualifying for CR, ie, both neutrophil >=0.5*10^9/L and platelets >=50*10^9/L must be met, but does not satisfy both neutrophils >=1*10^9/L and platelets >=100*10^9/L at the same time; absence of extramedullary disease; and absence of blasts with Auer rods.
Time Frame: From the date of randomization to the first documentation of response (CRi/CRh or better) (maximum up to 3 years)
Population: FA set included all randomized participants.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Non-intensive Study: Glasdegib + Azacitidine | Non-intensive Study: Placebo + Azacitidine
Number analyzed (Participants) | 163 | 162
Months
  TTRi | 4.057 (1.9532) | 4.093 (2.1809)
  TTRh | 4.334 (1.8853) | 4.146 (2.1540)

19. Secondary Outcome: Intensive Study: Event-free Survival (EFS)
Description: EFS: Time from the date of randomization to the date of treatment failure (TF), relapse from CR, or death from any cause, whichever comes first. TF was defined as failure to achieve CR during the induction cycle (including the re-induction cycle if there is one) and the event date for TF is the day of randomization. CR was defined based on 2017 ELN recommendations. CR: Bone marrow blasts <5%; absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease; ANC >=1.0*10^9/L; platelet count >=100*10^9/L.
Time Frame: From the date of randomization to the date of TF, relapse from CR, or death from any cause, whichever comes first (maximum up to 2 years)
Population: The intensive cohort was terminated because of futility. Participants ended study intervention early and were not followed up as planned. Hence, EFS was not collected, analyzed and reported.
Arm/Group | Intensive Study: Glasdegib + Cytarabine + Daunorubicin | Intensive Study: Placebo + Cytarabine + Daunorubicin
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Non-intensive Study: Event-free Survival (EFS)
Description: EFS: Time from the date of randomization to the date of TF, relapse from CR, or death from any cause, whichever comes first. TF was defined as failure to achieve CR during the induction cycle (including the re-induction cycle if there is one) and the event date for TF is the day of randomization. CR was defined based on 2017 ELN recommendations. CR: Bone marrow blasts <5%; absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease; ANC >=1.0*10^9/L; platelet count >=100*10^9/L.
Time Frame: From the date of randomization to the date of TF, relapse from CR, or death from any cause, whichever comes first (maximum up to 3 years)
Population: The non-intensive cohort was terminated because of futility. Participants ended study intervention early and were not followed up as planned. Hence, EFS was not collected, analyzed and reported.
Arm/Group | Non-intensive Study: Glasdegib + Azacitidine | Non-intensive Study: Placebo + Azacitidine
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Intensive Study: MD Anderson Symptom Inventory -Acute Myelogenous Leukemia/Myelodysplastic Syndrome (MDASI-AML/MDS) Score
Description: MDASI-AML/MDS: consists of 23 items, 13-item core cancer symptoms (pain, fatigue, nausea, disturbed sleep, distress, shortness of breath, problem remembering, lack of appetite, drowsiness, dry mouth, sadness, vomiting, and numbness), 4-item AML/MDS specific symptoms (malaise, diarrhea, muscle weakness, and skin problems), and 6 areas of interference (general activity, mood, work, walking, relations with other people, and enjoyment of life). The 13 core symptoms and 6 core interference items had highest frequency and/or severity in participants with various cancers and treatment types. It was measured at severity of symptoms and related interference at their worst level in last 24 hours by asking participants to respond to each item on an 0-10 NRS, where 0 = "not present" or "did not interfere" and 10 = "worst" or "interfered completely".
Time Frame: Day 1 up to maximum of 2 years
Population: The intensive cohort was terminated because of futility. Participants ended study intervention early and were not followed up as planned. Hence, MDASI-AML/MDS was not collected, analyzed and reported.
Arm/Group | Intensive Study: Glasdegib + Cytarabine + Daunorubicin | Intensive Study: Placebo + Cytarabine + Daunorubicin
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Non-intensive Study: MD Anderson Symptom Inventory -Acute Myelogenous Leukemia/Myelodysplastic Syndrome (MDASI-AML/MDS) Score
Description: as for outcome 21
Time Frame: Day 1 up to maximum of 3 years
Population: The non-intensive cohort was terminated because of futility. Participants ended study intervention early and were not followed up as planned. Hence, MDASI-AML/MDS was not collected, analyzed and reported.
Arm/Group | Non-intensive Study: Glasdegib + Azacitidine | Non-intensive Study: Placebo + Azacitidine
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Intensive Study: EuroQoL 5 Dimension Questionnaire 5-Level Version (EQ-5D-5L) Score
Description: EQ-5D-5L: brief, self-administered, validated and reliable generic health status instrument developed by the EuroQoL Group. It consists of the EQ-5D descriptive system and a visual analogue scale (VAS), the EuroQoL visual analogue scale (EQ-VAS). EQ-5D: descriptive system measures a participant's health state on 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Participant is asked to indicate his/her health state by rating each dimension on a 5-level scale (1=no problem, 5=extreme problem). This rating resulted in a 1-digit number expressing the level selected for that dimension. The digits for the 5 dimensions were combined in a 5-digit number describing the respondent's health state. The EQ-5D index scores ranges from 0 to 1, with 0=worst health state and 1=perfect health.
Time Frame: Day 1 up to maximum of 2 years
Population: The intensive cohort was terminated because of futility. Participants ended study intervention early and were not followed up as planned. Hence, EQ-5D-5L was not collected, analyzed and reported.
Arm/Group | Intensive Study: Glasdegib + Cytarabine + Daunorubicin | Intensive Study: Placebo + Cytarabine + Daunorubicin
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Non-intensive Study: EuroQoL 5 Dimension Questionnaire 5-Level Version (EQ-5D-5L) Score
Description: EQ-5D-5L: brief, self-administered, validated and reliable generic health status instrument developed by the EuroQoL group. It consists of the EQ-5D descriptive system and a VAS, EQ-VAS. EQ-5D: descriptive system measures a participant's health state on 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Participant is asked to indicate his/her health state by rating each dimension on a 5-level scale (1=no problem, 5=extreme problem). This rating resulted in a 1-digit number expressing the level selected for that dimension. The digits for the 5 dimensions were combined in a 5-digit number describing the respondent's health state. The EQ-5D index scores ranges from 0 to 1, with 0=worst health state and 1=perfect health.
Time Frame: Day 1 up to maximum of 3 years
Population: The non-intensive cohort was terminated because of futility. Participants ended study intervention early and were not followed up as planned. Hence, EQ-5D-5L was not collected, analyzed and reported.
Arm/Group | Non-intensive Study: Glasdegib + Azacitidine | Non-intensive Study: Placebo + Azacitidine
Number analyzed (Participants) | 0 | 0

25. Secondary Outcome: Intensive Study: EuroQoL Visual Analogue Scale (EQ-VAS)
Description: EQ-5D-5L: brief, self-administered, validated and reliable generic health status instrument developed by the EuroQoL group. It consists of the EQ-5D descriptive system and a VAS, EQ-VAS. EQ VAS records the respondent's self-rated health on a 20-cm vertical, VAS from 0 (worst imaginable health state) to 100 (best imaginable health state).
Time Frame: Day 1 up to maximum of 2 years
Population: The intensive cohort was terminated because of futility. Participants ended study intervention early and were not followed up as planned. Hence, EQ-VAS was not collected, analyzed and reported.
Arm/Group | Intensive Study: Glasdegib + Cytarabine + Daunorubicin | Intensive Study: Placebo + Cytarabine + Daunorubicin
Number analyzed (Participants) | 0 | 0

26. Secondary Outcome: Non-intensive Study: EuroQoL Visual Analogue Scale (EQ-VAS)
Description: as for outcome 25
Time Frame: Day 1 up to maximum of 3 years
Population: The non-intensive cohort was terminated because of futility. Participants ended study intervention early and were not followed up as planned. Hence, EQ-VAS was not collected, analyzed and reported.
Arm/Group | Non-intensive Study: Glasdegib + Azacitidine | Non-intensive Study: Placebo + Azacitidine
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: Intensive Study: Participants Global Impression of Symptoms (PGIS)
Description: PGIS: is a single 1-item questionnaire designed to assess participant's overall impression of disease severity at a given point in time. It uses a 4-point Likert scale as follows: In the last 24 hours, symptoms are: 1-"absent (no symptoms)", 2-"mild", 3-" moderate", 4="severe".
Time Frame: Day 1 up to maximum of 2 years
Population: The intensive cohort was terminated because of futility. Participants ended study intervention early and were not followed up as planned. Hence, PGIS was not collected, analyzed and reported.
Arm/Group | Intensive Study: Glasdegib + Cytarabine + Daunorubicin | Intensive Study: Placebo + Cytarabine + Daunorubicin
Number analyzed (Participants) | 0 | 0

28. Secondary Outcome: Non-intensive Study: Participants Global Impression of Symptoms (PGIS)
Description: as for outcome 27
Time Frame: Day 1 up to maximum of 3 years
Population: The non-intensive cohort was terminated because of futility. Participants ended study intervention early and were not followed up as planned. Hence, PGIS was not collected, analyzed and reported.
Arm/Group | Non-intensive Study: Glasdegib + Azacitidine | Non-intensive Study: Placebo + Azacitidine
Number analyzed (Participants) | 0 | 0

29. Secondary Outcome: Intensive Study: Participants Global Impression of Change (PGIC)
Description: PGIC: a single-item questionnaire designed to assess the participant's overall sense of whether there has been a change since starting treatment as rated on a 7-point Likert scale anchored by (1) 'very much improved' to (7) 'very much worse', with (4) =' no change'. The PGIC is a measure of "participant rating of global improvement and satisfaction with treatment".
Time Frame: Day 1 up to maximum of 2 years
Population: The intensive cohort was terminated because of futility. Participants ended study intervention early and were not followed up as planned. Hence, PGIC was not collected, analyzed and reported.
Arm/Group | Intensive Study: Glasdegib + Cytarabine + Daunorubicin | Intensive Study: Placebo + Cytarabine + Daunorubicin
Number analyzed (Participants) | 0 | 0

30. Secondary Outcome: Non-intensive Study: Participants Global Impression of Change (PGIC)
Description: as for outcome 29
Time Frame: Day 1 up to maximum of 3 years
Population: The non-intensive cohort was terminated because of futility. Participants ended study intervention early and were not followed up as planned. Hence, PGIC was not collected, analyzed and reported.
Arm/Group | Non-intensive Study: Glasdegib + Azacitidine | Non-intensive Study: Placebo + Azacitidine
Number analyzed (Participants) | 0 | 0

31. Secondary Outcome: Intensive Study: Number of Participants With Adverse Events (AEs),Serious Adverse Events (SAEs) and According to Severity AEs Graded by NCI CTCAE v.4.03
Description: AE: any untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship. SAE: any AE, regardless of dose, that led to death; was life-threatening; required hospitalization or prolonged hospitalization; led to persistent or significant incapacity or led to congenital anomaly or birth defect. AEs included SAEs and all non-SAEs. NCI CTCAE v.4.03, Grade 3=severe adverse event, Grade 4= life threatening consequences; urgent intervention indicated, Grade 5= death related to adverse event.
Time Frame: Day 1 up to maximum of 2 years
Population: Safety Analysis (SA) set included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive Study: Glasdegib + Cytarabine + Daunorubicin | Intensive Study: Placebo + Cytarabine + Daunorubicin
Number analyzed (Participants) | 198 | 201
Participants
  AEs | 196 | 198
  SAEs | 86 | 92
  Grade 3 or 4 AE | 173 | 169
  Grade 5 AE | 16 | 20

32. Secondary Outcome: Non-intensive Study: Number of Participants With Adverse Events (AEs),Serious Adverse Events (SAEs) and According to Severity AEs Graded by NCI CTCAE v.4.03
Description: as for outcome 31
Time Frame: Day 1 up to maximum of 3 years
Population: SA set included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Non-intensive Study: Glasdegib + Azacitidine | Non-intensive Study: Placebo + Azacitidine
Number analyzed (Participants) | 162 | 160
Participants
  AEs | 161 | 158
  SAEs | 117 | 124
  Grade 3 or 4 AE | 106 | 100
  Grade 5 AE | 50 | 52

33. Secondary Outcome: Intensive Study: Number of Participants With Treatment Related Adverse Events (AEs) and Serious Adverse Events (SAEs) Graded by NCI CTCAE v.4.03
Description: A treatment-related AE was any untoward medical occurrence attributed to the study drug in a participant who received study drug. SAE: any AE, regardless of dose, that led to death; was life-threatening; required hospitalization or prolonged hospitalization; led to persistent or significant incapacity or led to congenital anomaly or birth defect. NCI CTCAE v.4.03, Grade 3=severe adverse event, Grade 4= life threatening consequences; urgent intervention indicated, Grade 5= death related to adverse event.
Time Frame: Day 1 up to maximum of 2 years
Population: SA set included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive Study: Glasdegib + Cytarabine + Daunorubicin | Intensive Study: Placebo + Cytarabine + Daunorubicin
Number analyzed (Participants) | 198 | 201
Participants
  Treatment related AEs | 181 | 188
  Treatment related SAEs | 48 | 60
  Grade 3 or 4 AE | 161 | 149
  Grade 5 AE | 5 | 8

34. Secondary Outcome: Non-intensive Study: Number of Participants With Treatment Related Adverse Events (AEs) and Serious Adverse Events (SAEs) Graded by NCI CTCAE v.4.03
Description: A treatment-related AE was any untoward medical occurrence attributed to the study drug in a participant who received study drug. SAE: any AE, regardless of dose, that led to death; was life-threatening; required hospitalization or prolonged hospitalization; led to persistent or significant incapacity or led to congenital anomaly or birth defect. NCI CTCAE v4.03, Grade 3=severe adverse event, Grade 4= life threatening consequences; urgent intervention indicated, Grade 5= death related to adverse event.
Time Frame: Day 1 up to maximum of 3 years
Population: SA set included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Non-intensive Study: Glasdegib + Azacitidine | Non-intensive Study: Placebo + Azacitidine
Number analyzed (Participants) | 162 | 160
Participants
  Treatment related AEs | 133 | 123
  Treatment related SAEs | 45 | 37
  Grade 3 or 4 AE | 97 | 72
  Grade 5 AE | 4 | 4

35. Secondary Outcome: Intensive Study: Number of Participants With Shift From Baseline in Hematological Laboratory Abnormalities Graded by NCI CTCAE v.4.03
Description: Hematology laboratory test included: anemia, hemoglobin increased, international normalized ratio (INR) increased, lymphocyte count decreased, lymphocyte count increased, neutrophil count decreased, platelet count decreased, and white blood cell decreased. Laboratory results were categorically summarized according to the NCI-CTCAE criteria v4.03. Grade 1= mild; Grade 2= moderate; Grade 3= severe and Grade 4= life-threatening or disabling. Number of participants with shift from baseline for hematology laboratory test were assessed. Only those laboratory test parameters in which at least 1 participant had data were reported.
Time Frame: Day 1 up to maximum of 2 years
Population: SA set included all participants who received at least one dose of study drug. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "Number Analyzed" signifies participants evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive Study: Glasdegib + Cytarabine + Daunorubicin | Intensive Study: Placebo + Cytarabine + Daunorubicin
Number analyzed (Participants) | 196 | 197
Participants
  Anemia: Missing (baseline grade) to Grade 3/4 (CTCAE grade) | 0 | 2
  Anemia: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 27 | 14
  Anemia: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 113 | 103
  Anemia: Grade 3/4 (baseline grade) to Grade <=2 (CTCAE grade) | 4 | 5
  Anemia: Grade 3/4 (baseline grade) to Grade 3/4 (CTCAE grade) | 52 | 73
  Hemoglobin increased: Missing (baseline grade) to Grade <=2 (CTCAE grade) | 0 | 2
  Hemoglobin increased: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 194 | 194
  Hemoglobin increased: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 2 | 1
  INR increased: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 3 | 1
  INR increased: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 3 | 1
  Lymphocyte count decreased: Missing (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 193 | 193
  Lymphocyte count decreased: Missing (baseline grade) to Grade <=2 (CTCAE grade) | 0 | 2
  Lymphocyte count decreased: Missing (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 193 | 193
  Lymphocyte count decreased: Missing (baseline grade) to Grade 3/4 (CTCAE grade) | 0 | 4
  Lymphocyte count decreased: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 193 | 193
  Lymphocyte count decreased: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 21 | 26
  Lymphocyte count decreased: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 193 | 193
  Lymphocyte count decreased: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 160 | 152
  Lymphocyte count decreased: Grade 3/4 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 193 | 193
  Lymphocyte count decreased: Grade 3/4 (baseline grade) to Grade <=2 (CTCAE grade) | 1 | 0
  Lymphocyte count decreased: Grade 3/4 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 193 | 193
  Lymphocyte count decreased: Grade 3/4 (baseline grade) to Grade 3/4 (CTCAE grade) | 11 | 9
  Lymphocyte count increased: Missing (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 193 | 193
  Lymphocyte count increased: Missing (baseline grade) to Grade <=2 (CTCAE grade) | 0 | 6
  Lymphocyte count increased: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 193 | 193
  Lymphocyte count increased: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 185 | 180
  Lymphocyte count increased: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 193 | 193
  Lymphocyte count increased: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 6 | 4
  Lymphocyte count increased: Grade 3/4 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 193 | 193
  Lymphocyte count increased: Grade 3/4 (baseline grade) to Grade <=2 (CTCAE grade) | 1 | 3
  Lymphocyte count increased: Grade 3/4 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 193 | 193
  Lymphocyte count increased: Grade 3/4 (baseline grade) to Grade 3/4 (CTCAE grade) | 1 | 0
  Neutrophil count decreased: Missing (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 194 | 193
  Neutrophil count decreased: Missing (baseline grade) to Grade 3/4 (CTCAE grade) | 0 | 4
  Neutrophil count decreased: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 194 | 193
  Neutrophil count decreased: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 4 | 2
  Neutrophil count decreased: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 194 | 193
  Neutrophil count decreased: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 85 | 79
  Neutrophil count decreased: Grade 3/4 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 194 | 193
  Neutrophil count decreased: Grade 3/4 (baseline grade) to Grade <=2 (CTCAE grade) | 0 | 2
  Neutrophil count decreased: Grade 3/4 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 194 | 193
  Neutrophil count decreased: Grade 3/4 (baseline grade) to Grade 3/4 (CTCAE grade) | 105 | 106
  Platelet count decreased: Missing (baseline grade) to Grade 3/4 (CTCAE grade) | 1 | 2
  Platelet count decreased: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 98 | 100
  Platelet count decreased: Grade 3/4 (baseline grade) to Grade 3/4 (CTCAE grade) | 97 | 95
  White blood cell decreased: Missing (baseline grade) to Grade 3/4 (CTCAE grade) | 1 | 4
  White blood cell decreased: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 3 | 2
  White blood cell decreased: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 155 | 156
  White blood cell decreased: Grade 3/4 (baseline grade) to Grade 3/4 (CTCAE grade) | 37 | 35

36. Secondary Outcome: Non-intensive Study: Number of Participants With Shift From Baseline in Hematological Laboratory Abnormalities Graded by NCI CTCAE v.4.03
Description: Hematology laboratory test included: anemia, hemoglobin increased, INR increased, lymphocyte count decreased, lymphocyte count increased, neutrophil count decreased, platelet count decreased, and white blood cell decreased. Laboratory results were categorically summarized according to the NCI-CTCAE criteria v4.03. Grade 1= mild; Grade 2= moderate; Grade 3= severe and Grade 4= life-threatening or disabling. Number of participants with shift from baseline for hematology laboratory test were assessed. Only those laboratory test parameters in which at least 1 participant had data were reported.
Time Frame: Day 1 up to maximum of 3 years
Population: as for outcome 35
Measure: Count of Participants; unit: Participants
Arm/Group | Non-intensive Study: Glasdegib + Azacitidine | Non-intensive Study: Placebo + Azacitidine
Number analyzed (Participants) | 162 | 160
Participants
  Anemia: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 160 | 160
  Anemia: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 29 | 41
  Anemia: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 160 | 160
  Anemia: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 97 | 87
  Anemia: Grade 3/4 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 160 | 160
  Anemia: Grade 3/4 (baseline grade) to Grade <=2 (CTCAE grade) | 5 | 1
  Anemia: Grade 3/4 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 160 | 160
  Anemia: Grade 3/4 (baseline grade) to Grade 3/4 (CTCAE grade) | 29 | 31
  Hemoglobin increased: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 160 | 160
  Hemoglobin increased: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 160 | 159
  Hemoglobin increased: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 160 | 160
  Hemoglobin increased: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 0 | 1
  Lymphocyte count decreased: Missing (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 159 | 160
  Lymphocyte count decreased: Missing (baseline grade) to Grade <=2 (CTCAE grade) | 2 | 0
  Lymphocyte count decreased: Missing (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 159 | 160
  Lymphocyte count decreased: Missing (baseline grade) to Grade 3/4 (CTCAE grade) | 1 | 0
  Lymphocyte count decreased: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 159 | 160
  Lymphocyte count decreased: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 96 | 89
  Lymphocyte count decreased: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 159 | 160
  Lymphocyte count decreased: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 51 | 54
  Lymphocyte count decreased: Grade 3/4 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 159 | 160
  Lymphocyte count decreased: Grade 3/4 (baseline grade) to Grade <=2 (CTCAE grade) | 2 | 4
  Lymphocyte count decreased: Grade 3/4 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 159 | 160
  Lymphocyte count decreased: Grade 3/4 (baseline grade) to Grade 3/4 (CTCAE grade) | 7 | 13
  Lymphocyte count increased: Missing (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 159 | 160
  Lymphocyte count increased: Missing (baseline grade) to Grade <=2 (CTCAE grade) | 3 | 0
  Lymphocyte count increased: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 159 | 160
  Lymphocyte count increased: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 147 | 157
  Lymphocyte count increased: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 159 | 160
  Lymphocyte count increased: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 7 | 3
  Lymphocyte count increased: Grade 3/4 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 159 | 160
  Lymphocyte count increased: Grade 3/4 (baseline grade) to Grade 3/4 (CTCAE grade) | 2 | 0
  Neutrophil count decreased: Missing (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 159 | 160
  Neutrophil count decreased: Missing (baseline grade) to Grade 3/4 (CTCAE grade) | 4 | 0
  Neutrophil count decreased: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 159 | 160
  Neutrophil count decreased: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 13 | 22
  Neutrophil count decreased: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 159 | 160
  Neutrophil count decreased: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 48 | 40
  Neutrophil count decreased: Grade 3/4 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 159 | 160
  Neutrophil count decreased: Grade 3/4 (baseline grade) to Grade <=2 (CTCAE grade) | 2 | 1
  Neutrophil count decreased: Grade 3/4 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 159 | 160
  Neutrophil count decreased: Grade 3/4 (baseline grade) to Grade 3/4 (CTCAE grade) | 92 | 97
  Platelet count decreased: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 160 | 160
  Platelet count decreased: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 21 | 28
  Platelet count decreased: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 160 | 160
  Platelet count decreased: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 55 | 64
  Platelet count decreased: Grade 3/4 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 160 | 160
  Platelet count decreased: Grade 3/4 (baseline grade) to Grade <=2 (CTCAE grade) | 1 | 0
  Platelet count decreased: Grade 3/4 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 160 | 160
  Platelet count decreased: Grade 3/4 (baseline grade) to Grade 3/4 (CTCAE grade) | 83 | 68
  White blood cell decreased: Missing (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 160 | 159
  White blood cell decreased: Missing (baseline grade) to Grade <=2 (CTCAE grade) | 1 | 0
  White blood cell decreased: Missing (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 160 | 159
  White blood cell decreased: Missing (baseline grade) to Grade 3/4 (CTCAE grade) | 1 | 0
  White blood cell decreased: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 160 | 159
  White blood cell decreased: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 43 | 48
  White blood cell decreased: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 160 | 159
  White blood cell decreased: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 70 | 62
  White blood cell decreased: Grade 3/4 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 160 | 159
  White blood cell decreased: Grade 3/4 (baseline grade) to Grade <=2 (CTCAE grade) | 0 | 1
  White blood cell decreased: Grade 3/4 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 160 | 159
  White blood cell decreased: Grade 3/4 (baseline grade) to Grade 3/4 (CTCAE grade) | 45 | 48

37. Secondary Outcome: Intensive Study: Number of Participants With Shift From Baseline in Chemistry Laboratory Abnormalities Graded by NCI CTCAE v.4.03
Description: Chemistry laboratory test included: alanine aminotransferase increased, alkaline phosphatase increased, aspartate aminotransferase increased, blood bilirubin increased, chronic kidney disease, creatine phosphokinase (CPK) increased, creatinine increased, gamma glutamyl transferase (GGT) increased, hypercalcemia, hyperglycemia, hyperkalemia, hypermagnesemia, hypernatremia, hypoalbuminemia, hypocalcemia, hypoglycemia, hypokalemia, hypomagnesemia, hyponatremia, and hypophosphatemia. Laboratory results were categorically summarized according to the NCI-CTCAE criteria v4.03. Grade 1= mild; Grade 2= moderate; Grade 3= severe and Grade 4= life-threatening or disabling. Number of participants with shift from baseline for chemistry laboratory test were assessed. Only those laboratory test parameters in which at least 1 participant had data were reported.
Time Frame: Day 1 up to maximum of 2 years
Population: SA set included all participants who received at least one dose of study drug. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "Number Analyzed" signifies participants evaluable for specific rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive Study: Glasdegib + Cytarabine + Daunorubicin | Intensive Study: Placebo + Cytarabine + Daunorubicin
Number analyzed (Participants) | 196 | 198
Participants
  Alanine aminotransferase increased: Missing (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 193 | 198
  Alanine aminotransferase increased: Missing (baseline grade) to Grade <=2 (CTCAE grade) | 1 | 1
  Alanine aminotransferase increased: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 193 | 198
  Alanine aminotransferase increased: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 175 | 184
  Alanine aminotransferase increased: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 193 | 198
  Alanine aminotransferase increased: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 16 | 13
  Alanine aminotransferase increased: Grade 3/4 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 193 | 198
  Alanine aminotransferase increased: Grade 3/4 (baseline grade) to Grade <=2 (CTCAE grade) | 1 | 0
  Alkaline phosphatase increased: Missing (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 191 | 198
  Alkaline phosphatase increased: Missing (baseline grade) to Grade <=2 (CTCAE grade) | 2 | 3
  Alkaline phosphatase increased: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 191 | 198
  Alkaline phosphatase increased: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 187 | 192
  Alkaline phosphatase increased: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 191 | 198
  Alkaline phosphatase increased: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 2 | 3
  Aspartate aminotransferase increased: Missing (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 193 | 198
  Aspartate aminotransferase increased: Missing (baseline grade) to Grade <=2 (CTCAE grade) | 5 | 2
  Aspartate aminotransferase increased: Missing (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 193 | 198
  Aspartate aminotransferase increased: Missing (baseline grade) to Grade 3/4 (CTCAE grade) | 0 | 1
  Aspartate aminotransferase increased: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 193 | 198
  Aspartate aminotransferase increased: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 173 | 186
  Aspartate aminotransferase increased: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 193 | 198
  Aspartate aminotransferase increased: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 15 | 9
  Blood bilirubin increased: Missing (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 192 | 198
  Blood bilirubin increased: Missing (baseline grade) to Grade <=2 (CTCAE grade) | 0 | 3
  Blood bilirubin increased: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 192 | 198
  Blood bilirubin increased: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 184 | 189
  Blood bilirubin increased: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 192 | 198
  Blood bilirubin increased: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 8 | 5
  Blood bilirubin increased: Grade 3/4 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 192 | 198
  Blood bilirubin increased: Grade 3/4 (baseline grade) to Grade 3/4 (CTCAE grade) | 0 | 1
  Chronic kidney disease: Missing (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 195 | 198
  Chronic kidney disease: Missing (baseline grade) to Grade <=2 (CTCAE grade) | 4 | 5
  Chronic kidney disease: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 195 | 198
  Chronic kidney disease: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 182 | 188
  Chronic kidney disease: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 195 | 198
  Chronic kidney disease: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 8 | 4
  Chronic kidney disease: Grade 3/4 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 195 | 198
  Chronic kidney disease: Grade 3/4 (baseline grade) to Grade <=2 (CTCAE grade) | 1 | 0
  Chronic kidney disease: Grade 3/4 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 195 | 198
  Chronic kidney disease: Grade 3/4 (baseline grade) to Grade 3/4 (CTCAE grade) | 0 | 1
  CPK increased: Missing (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 183 | 185
  CPK increased: Missing (baseline grade) to Grade <=2 (CTCAE grade) | 20 | 19
  CPK increased: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 183 | 185
  CPK increased: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 161 | 166
  CPK increased: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 183 | 185
  CPK increased: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 2 | 0
  Creatinine increased: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 195 | 198
  Creatinine increased: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 188 | 192
  Creatinine increased: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 195 | 198
  Creatinine increased: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 7 | 6
  GGT increased: Missing (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 13 | 20
  GGT increased: Missing (baseline grade) to Grade <=2 (CTCAE grade) | 5 | 7
  GGT increased: Missing (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 13 | 20
  GGT increased: Missing (baseline grade) to Grade 3/4 (CTCAE grade) | 8 | 11
  GGT increased: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 13 | 20
  GGT increased: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 0 | 2
  Hypercalcemia: Missing (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 192 | 197
  Hypercalcemia: Missing (baseline grade) to Grade <=2 (CTCAE grade) | 1 | 5
  Hypercalcemia: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 192 | 197
  Hypercalcemia: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 191 | 192
  Hyperglycemia: Missing (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 194 | 198
  Hyperglycemia: Missing (baseline grade) to Grade <=2 (CTCAE grade) | 1 | 3
  Hyperglycemia: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 194 | 198
  Hyperglycemia: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 174 | 183
  Hyperglycemia: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 194 | 198
  Hyperglycemia: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 15 | 10
  Hyperglycemia: Grade 3/4 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 194 | 198
  Hyperglycemia: Grade 3/4 (baseline grade) to Grade <=2 (CTCAE grade) | 2 | 1
  Hyperglycemia: Grade 3/4 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 194 | 198
  Hyperglycemia: Grade 3/4 (baseline grade) to Grade 3/4 (CTCAE grade) | 2 | 1
  Hyperkalemia: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 194 | 194
  Hyperkalemia: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 2 | 3
  Hyperkalemia: Grade 3/4 (baseline grade) to Grade <=2 (CTCAE grade) | 0 | 1
  Hypermagnesemia: Missing (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 193 | 192
  Hypermagnesemia: Missing (baseline grade) to Grade <=2 (CTCAE grade) | 2 | 4
  Hypermagnesemia: Missing (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 193 | 192
  Hypermagnesemia: Missing (baseline grade) to Grade 3/4 (CTCAE grade) | 0 | 1
  Hypermagnesemia: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 193 | 192
  Hypermagnesemia: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 190 | 184
  Hypermagnesemia: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 193 | 192
  Hypermagnesemia: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 1 | 2
  Hypermagnesemia: Grade 3/4 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 193 | 192
  Hypermagnesemia: Grade 3/4 (baseline grade) to Grade <=2 (CTCAE grade) | 0 | 1
  Hypernatremia: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 196 | 196
  Hypernatremia: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 0 | 1
  Hypernatremia: Grade 3/4 (baseline grade) to Grade <=2 (CTCAE grade) | 0 | 1
  Hypoalbuminemia: Missing (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 192 | 198
  Hypoalbuminemia: Missing (baseline grade) to Grade <=2 (CTCAE grade) | 0 | 3
  Hypoalbuminemia: Missing (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 192 | 198
  Hypoalbuminemia: Missing (baseline grade) to Grade 3/4 (CTCAE grade) | 1 | 1
  Hypoalbuminemia: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 192 | 198
  Hypoalbuminemia: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 185 | 185
  Hypoalbuminemia: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 192 | 198
  Hypoalbuminemia: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 5 | 8
  Hypoalbuminemia: Grade 3/4 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 192 | 198
  Hypoalbuminemia: Grade 3/4 (baseline grade) to Grade 3/4 (CTCAE grade) | 1 | 1
  Hypocalcemia: Missing (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 192 | 197
  Hypocalcemia: Missing (baseline grade) to Grade <=2 (CTCAE grade) | 1 | 5
  Hypocalcemia: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 192 | 197
  Hypocalcemia: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 190 | 189
  Hypocalcemia: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 192 | 197
  Hypocalcemia: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 1 | 3
  Hypoglycemia: Missing (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 194 | 198
  Hypoglycemia: Missing (baseline grade) to Grade <=2 (CTCAE grade) | 1 | 3
  Hypoglycemia: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 194 | 198
  Hypoglycemia: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 193 | 194
  Hypoglycemia: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 194 | 198
  Hypoglycemia: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 0 | 1
  Hypokalemia: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 155 | 159
  Hypokalemia: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 41 | 37
  Hypokalemia: Grade 3/4 (baseline grade) to Grade <=2 (CTCAE grade) | 0 | 2
  Hypomagnesemia: Missing (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 193 | 192
  Hypomagnesemia: Missing (baseline grade) to Grade <=2 (CTCAE grade) | 2 | 5
  Hypomagnesemia: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 193 | 192
  Hypomagnesemia: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 190 | 187
  Hypomagnesemia: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 193 | 192
  Hypomagnesemia: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 1 | 0
  Hyponatremia: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 177 | 188
  Hyponatremia: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 17 | 8
  Hyponatremia: Grade 3/4 (baseline grade) to Grade <=2 (CTCAE grade) | 1 | 1
  Hyponatremia: Grade 3/4 (baseline grade) to Grade 3/4 (CTCAE grade) | 1 | 1
  Hypophosphatemia: Missing (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 193 | 193
  Hypophosphatemia: Missing (baseline grade) to Grade <=2 (CTCAE grade) | 3 | 3
  Hypophosphatemia: Missing (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 193 | 193
  Hypophosphatemia: Missing (baseline grade) to Grade 3/4 (CTCAE grade) | 1 | 1
  Hypophosphatemia: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 193 | 193
  Hypophosphatemia: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 153 | 153
  Hypophosphatemia: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade: number analyzed (Participants) | 193 | 193
  Hypophosphatemia: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade | 33 | 33
  Hypophosphatemia: Grade 3/4 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 193 | 193
  Hypophosphatemia: Grade 3/4 (baseline grade) to Grade <=2 (CTCAE grade) | 0 | 2
  Hypophosphatemia: Grade 3/4 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 193 | 193
  Hypophosphatemia: Grade 3/4 (baseline grade) to Grade 3/4 (CTCAE grade) | 3 | 1

38. Secondary Outcome: Non-intensive Study: Number of Participants With Shift From Baseline in Chemistry Laboratory Abnormalities Graded by NCI CTCAE v.4.03
Description: Chemistry laboratory test included: alanine aminotransferase increased, alkaline phosphatase increased, aspartate aminotransferase increased, blood bilirubin increased, chronic kidney disease, CPK increased, creatinine increased, GGT increased, hypercalcemia, hyperglycemia, hyperkalemia, hypermagnesemia, hypernatremia, hypoalbuminemia, hypocalcemia, hypoglycemia, hypokalemia, hypomagnesemia, hyponatremia, and hypophosphatemia. Laboratory results were categorically summarized according to the NCI-CTCAE criteria v4.03. Grade 1= mild; Grade 2= moderate; Grade 3= severe and Grade 4= life-threatening or disabling. Number of participants with shift from baseline for chemistry laboratory test were assessed. Only those laboratory test parameters in which at least 1 participant had data were reported.
Time Frame: Day 1 up to maximum of 3 years
Population: as for outcome 37
Measure: Count of Participants; unit: Participants
Arm/Group | Non-intensive Study: Glasdegib + Azacitidine | Non-intensive Study: Placebo + Azacitidine
Number analyzed (Participants) | 160 | 160
Participants
  Alanine aminotransferase increased: Missing (baseline grade) to Grade <=2 (CTCAE grade) | 2 | 0
  Alanine aminotransferase increased: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 152 | 154
  Alanine aminotransferase increased: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 6 | 6
  Alanine aminotransferase increased: Grade 3/4 (baseline grade) to Grade <=2 (CTCAE grade) | 0 | 0
  Alkaline phosphatase increased: Missing (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 159 | 159
  Alkaline phosphatase increased: Missing (baseline grade) to Grade <=2 (CTCAE grade) | 0 | 1
  Alkaline phosphatase increased: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 159 | 159
  Alkaline phosphatase increased: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 159 | 157
  Alkaline phosphatase increased: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 159 | 159
  Alkaline phosphatase increased: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 0 | 1
  Aspartate aminotransferase increased: Missing (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 159 | 160
  Aspartate aminotransferase increased: Missing (baseline grade) to Grade <=2 (CTCAE grade) | 3 | 0
  Aspartate aminotransferase increased: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 159 | 160
  Aspartate aminotransferase increased: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 152 | 156
  Aspartate aminotransferase increased: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 159 | 160
  Aspartate aminotransferase increased: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 4 | 4
  Blood bilirubin increased: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 157 | 159
  Blood bilirubin increased: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 3 | 1
  Chronic kidney disease: Missing (baseline grade) to Grade <=2 (CTCAE grade) | 2 | 1
  Chronic kidney disease: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 130 | 134
  Chronic kidney disease: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 28 | 23
  Chronic kidney disease: Grade 3/4 (baseline grade) to Grade 3/4 (CTCAE grade) | 0 | 2
  CPK increased: Missing (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 157 | 157
  CPK increased: Missing (baseline grade) to Grade <=2 (CTCAE grade) | 9 | 8
  CPK increased: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 157 | 157
  CPK increased: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 147 | 147
  CPK increased: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 157 | 157
  CPK increased: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 1 | 2
  Creatinine increased: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 153 | 155
  Creatinine increased: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 7 | 5
  GGT increased: Missing (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 8 | 8
  GGT increased: Missing (baseline grade) to Grade <=2 (CTCAE grade) | 3 | 5
  GGT increased: Missing (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 8 | 8
  GGT increased: Missing (baseline grade) to Grade 3/4 (CTCAE grade) | 4 | 3
  GGT increased: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 8 | 8
  GGT increased: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 1 | 0
  Hypercalcemia: Missing (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 158 | 160
  Hypercalcemia: Missing (baseline grade) to Grade <=2 (CTCAE grade) | 2 | 2
  Hypercalcemia: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 158 | 160
  Hypercalcemia: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 156 | 158
  Hyperglycemia: Missing (baseline grade) to Grade <=2 (CTCAE grade) | 2 | 4
  Hyperglycemia: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 147 | 136
  Hyperglycemia: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 8 | 14
  Hyperglycemia: Grade 3/4 (baseline grade) to Grade <=2 (CTCAE grade) | 2 | 2
  Hyperkalemia: Missing (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 159 | 160
  Hyperkalemia: Missing (baseline grade) to Grade <=2 (CTCAE grade) | 2 | 0
  Hyperkalemia: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 159 | 160
  Hyperkalemia: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 155 | 157
  Hyperkalemia: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 159 | 160
  Hyperkalemia: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 2 | 3
  Hyperkalemia: Grade 3/4 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 159 | 160
  Hyperkalemia: Grade 3/4 (baseline grade) to Grade <=2 (CTCAE grade) | 0 | 0
  Hyperkalemia: Grade 3/4 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 159 | 160
  Hyperkalemia: Grade 3/4 (baseline grade) to Grade 3/4 (CTCAE grade) | 0 | 0
  Hypermagnesemia: Missing (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 159 | 160
  Hypermagnesemia: Missing (baseline grade) to Grade <=2 (CTCAE grade) | 2 | 4
  Hypermagnesemia: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 159 | 160
  Hypermagnesemia: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 155 | 154
  Hypermagnesemia: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 159 | 160
  Hypermagnesemia: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 2 | 2
  Hypernatremia: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 158 | 159
  Hypernatremia: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 2 | 1
  Hypoalbuminemia: Missing (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 159 | 160
  Hypoalbuminemia: Missing (baseline grade) to Grade <=2 (CTCAE grade) | 2 | 0
  Hypoalbuminemia: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 159 | 160
  Hypoalbuminemia: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 151 | 157
  Hypoalbuminemia: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 159 | 160
  Hypoalbuminemia: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 6 | 3
  Hypocalcemia: Missing (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 158 | 160
  Hypocalcemia: Missing (baseline grade) to Grade <=2 (CTCAE grade) | 2 | 2
  Hypocalcemia: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 158 | 160
  Hypocalcemia: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 154 | 155
  Hypocalcemia: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 158 | 160
  Hypocalcemia: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 1 | 3
  Hypocalcemia: Grade 3/4 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 158 | 160
  Hypocalcemia: Grade 3/4 (baseline grade) to Grade 3/4 (CTCAE grade) | 0 | 0
  Hypoglycemia: Missing (baseline grade) to Grade <=2 (CTCAE grade) | 2 | 4
  Hypoglycemia: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 155 | 156
  Hypoglycemia: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 3 | 0
  Hypokalemia: Missing (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 159 | 160
  Hypokalemia: Missing (baseline grade) to Grade <=2 (CTCAE grade) | 2 | 0
  Hypokalemia: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 159 | 160
  Hypokalemia: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 129 | 139
  Hypokalemia: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 159 | 160
  Hypokalemia: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 23 | 15
  Hypokalemia: Grade 3/4 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 159 | 160
  Hypokalemia: Grade 3/4 (baseline grade) to Grade <=2 (CTCAE grade) | 1 | 2
  Hypokalemia: Grade 3/4 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 159 | 160
  Hypokalemia: Grade 3/4 (baseline grade) to Grade 3/4 (CTCAE grade) | 4 | 4
  Hypomagnesemia: Missing (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 159 | 160
  Hypomagnesemia: Missing (baseline grade) to Grade <=2 (CTCAE grade) | 2 | 4
  Hypomagnesemia: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 159 | 160
  Hypomagnesemia: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 151 | 153
  Hypomagnesemia: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 159 | 160
  Hypomagnesemia: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 6 | 2
  Hypomagnesemia: Grade 3/4 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 159 | 160
  Hypomagnesemia: Grade 3/4 (baseline grade) to Grade <=2 (CTCAE grade) | 0 | 1
  Hyponatremia: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 135 | 142
  Hyponatremia: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade) | 24 | 15
  Hyponatremia: Grade 3/4 (baseline grade) to Grade <=2 (CTCAE grade) | 0 | 1
  Hyponatremia: Grade 3/4 (baseline grade) to Grade 3/4 (CTCAE grade) | 1 | 2
  Hypophosphatemia: Missing (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 158 | 160
  Hypophosphatemia: Missing (baseline grade) to Grade <=2 (CTCAE grade) | 3 | 2
  Hypophosphatemia: Missing (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 158 | 160
  Hypophosphatemia: Missing (baseline grade) to Grade 3/4 (CTCAE grade) | 1 | 0
  Hypophosphatemia: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 158 | 160
  Hypophosphatemia: Grade <=2 (baseline grade) to Grade <=2 (CTCAE grade) | 141 | 138
  Hypophosphatemia: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade: number analyzed (Participants) | 158 | 160
  Hypophosphatemia: Grade <=2 (baseline grade) to Grade 3/4 (CTCAE grade | 12 | 17
  Hypophosphatemia: Grade 3/4 (baseline grade) to Grade <=2 (CTCAE grade): number analyzed (Participants) | 158 | 160
  Hypophosphatemia: Grade 3/4 (baseline grade) to Grade <=2 (CTCAE grade) | 0 | 1
  Hypophosphatemia: Grade 3/4 (baseline grade) to Grade 3/4 (CTCAE grade): number analyzed (Participants) | 158 | 160
  Hypophosphatemia: Grade 3/4 (baseline grade) to Grade 3/4 (CTCAE grade) | 1 | 2

39. Secondary Outcome: Intensive Study: Number of Participants With Shift From Baseline in Coagulation Laboratory Abnormalities Graded by NCI CTCAE v.4.03
Description: Coagulation laboratory test included: activated partial thromboplastin time prolonged, and INR increased. Laboratory results were categorically summarized according to the NCI-CTCAE criteria v4.03. Grade 0= no abnormality; Grade 1= mild; Grade 2= moderate; Grade 3= severe and Grade 4= life-threatening or disabling. Number of participants with shift from baseline for coagulation were assessed. Only those laboratory test parameters in which at least 1 participant had data were reported.
Time Frame: Day 1 up to maximum of 2 years
Population: as for outcome 37
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive Study: Glasdegib + Cytarabine + Daunorubicin | Intensive Study: Placebo + Cytarabine + Daunorubicin
Number analyzed (Participants) | 6 | 11
Participants
  Activated partial thromboplastin time prolonged: Missing (baseline grade) to Grade 0 (CTCAE grade): number analyzed (Participants) | 4 | 9
  Activated partial thromboplastin time prolonged: Missing (baseline grade) to Grade 0 (CTCAE grade) | 1 | 0
  Activated partial thromboplastin time prolonged: Missing (baseline grade) to Grade 1 (CTCAE grade): number analyzed (Participants) | 4 | 9
  Activated partial thromboplastin time prolonged: Missing (baseline grade) to Grade 1 (CTCAE grade) | 0 | 1
  Activated partial thromboplastin time prolonged: Grade 0 (baseline grade) to Grade 0 (CTCAE grade): number analyzed (Participants) | 4 | 9
  Activated partial thromboplastin time prolonged: Grade 0 (baseline grade) to Grade 0 (CTCAE grade) | 0 | 4
  Activated partial thromboplastin time prolonged: Grade 0 (baseline grade) to Grade 1 (CTCAE grade): number analyzed (Participants) | 4 | 9
  Activated partial thromboplastin time prolonged: Grade 0 (baseline grade) to Grade 1 (CTCAE grade) | 1 | 2
  Activated partial thromboplastin time prolonged: Grade 0 (baseline grade) to Grade 2 (CTCAE grade): number analyzed (Participants) | 4 | 9
  Activated partial thromboplastin time prolonged: Grade 0 (baseline grade) to Grade 2 (CTCAE grade) | 0 | 1
  Activated partial thromboplastin time prolonged: Grade 0 (baseline grade) to Grade 3 (CTCAE grade): number analyzed (Participants) | 4 | 9
  Activated partial thromboplastin time prolonged: Grade 0 (baseline grade) to Grade 3 (CTCAE grade) | 1 | 0
  Activated partial thromboplastin time prolonged: Grade 1 (baseline grade) to Grade 1 (CTCAE grade): number analyzed (Participants) | 4 | 9
  Activated partial thromboplastin time prolonged: Grade 1 (baseline grade) to Grade 1 (CTCAE grade) | 1 | 1
  INR increased: Missing (baseline grade) to Grade 0 (CTCAE grade) | 1 | 1
  INR increased: Missing (baseline grade) to Grade 1 (CTCAE grade) | 0 | 1
  INR increased: Missing (baseline grade) to Grade 2 (CTCAE grade) | 1 | 0
  INR increased: Grade 0 (baseline grade) to Grade 0 (CTCAE grade) | 0 | 2
  INR increased: Grade 0 (baseline grade) to Grade 1 (CTCAE grade) | 1 | 0
  INR increased: Grade 0 (baseline grade) to Grade 2 (CTCAE grade) | 1 | 1
  INR increased: Grade 0 (baseline grade) to Grade 3 (CTCAE grade) | 0 | 1
  INR increased: Grade 1 (baseline grade) to Grade 0 (CTCAE grade) | 0 | 1
  INR increased: Grade 1 (baseline grade) to Grade 1 (CTCAE grade) | 0 | 3
  INR increased: Grade 1 (baseline grade) to Grade 2 (CTCAE grade) | 1 | 1
  INR increased: Grade 1 (baseline grade) to Grade 3 (CTCAE grade) | 1 | 0

40. Secondary Outcome: Non-intensive Study: Number of Participants With Shift From Baseline in Coagulation Laboratory Abnormalities Graded by NCI CTCAE v.4.03
Description: as for outcome 39
Time Frame: Day 1 up to maximum of 3 years
Population: as for outcome 37
Measure: Count of Participants; unit: Participants
Arm/Group | Non-intensive Study: Glasdegib + Azacitidine | Non-intensive Study: Placebo + Azacitidine
Number analyzed (Participants) | 17 | 13
Participants
  Activated partial thromboplastin time prolonged: Missing (baseline grade) to Grade 0 (CTCAE grade): number analyzed (Participants) | 17 | 12
  Activated partial thromboplastin time prolonged: Missing (baseline grade) to Grade 0 (CTCAE grade) | 1 | 0
  Activated partial thromboplastin time prolonged: Grade 0 (baseline grade) to Grade 0 (CTCAE grade): number analyzed (Participants) | 17 | 12
  Activated partial thromboplastin time prolonged: Grade 0 (baseline grade) to Grade 0 (CTCAE grade) | 8 | 5
  Activated partial thromboplastin time prolonged: Grade 0 (baseline grade) to Grade 1 (CTCAE grade): number analyzed (Participants) | 17 | 12
  Activated partial thromboplastin time prolonged: Grade 0 (baseline grade) to Grade 1 (CTCAE grade) | 5 | 7
  Activated partial thromboplastin time prolonged: Grade 1 (baseline grade) to Grade 0 (CTCAE grade): number analyzed (Participants) | 17 | 12
  Activated partial thromboplastin time prolonged: Grade 1 (baseline grade) to Grade 0 (CTCAE grade) | 1 | 0
  Activated partial thromboplastin time prolonged: Grade 1 (baseline grade) to Grade 1 (CTCAE grade): number analyzed (Participants) | 17 | 12
  Activated partial thromboplastin time prolonged: Grade 1 (baseline grade) to Grade 1 (CTCAE grade) | 1 | 0
  Activated partial thromboplastin time prolonged: Grade 2 (baseline grade) to Grade 1 (CTCAE grade): number analyzed (Participants) | 17 | 12
  Activated partial thromboplastin time prolonged: Grade 2 (baseline grade) to Grade 1 (CTCAE grade) | 1 | 0
  INR increased: Missing (baseline grade) to Grade 0 (CTCAE grade) | 1 | 0
  INR increased: Grade 0 (baseline grade) to Grade 0 (CTCAE grade) | 4 | 5
  INR increased: Grade 0 (baseline grade) to Grade 1 (CTCAE grade) | 6 | 4
  INR increased: Grade 0 (baseline grade) to Grade 2 (CTCAE grade) | 1 | 2
  INR increased: Grade 0 (baseline grade) to Grade 3 (CTCAE grade) | 1 | 0
  INR increased: Grade 1 (baseline grade) to Grade 1 (CTCAE grade) | 1 | 1
  INR increased: Grade 1 (baseline grade) to Grade 2 (CTCAE grade) | 2 | 0
  INR increased: Grade 3 (baseline grade) to Grade 1 (CTCAE grade) | 1 | 1

41. Secondary Outcome: Intensive Study: Plasma Trough Concentration (Ctrough) of Glasdegib
Description: Ctrough of Glasdegib was measured in nanogram per milliliter (ng/mL).
Time Frame: Induction, Day 10+/-1: pre-dose, 1, 4 hour (hr); Consolidation phase, Day 1: pre-dose, 1, 4 hr
Population: Analysis population included all participants who were treated and who had at least 1 value of analyte concentration of Glasdegib available. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "Number Analyzed" signifies participants evaluable for specific time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | Intensive Study: Glasdegib + Cytarabine + Daunorubicin
Number analyzed (Participants) | 123
ng/ml
  Induction Day 10: number analyzed (Participants) | 81
  Induction Day 10 | 413.54 (125)
  Consolidation 1, Day 1: number analyzed (Participants) | 33
  Consolidation 1, Day 1 | 245.48 (80)
  Consolidation 2, Day 1: number analyzed (Participants) | 41
  Consolidation 2, Day 1 | 259.79 (122)

42. Secondary Outcome: Non-intensive Study: Plasma Trough Concentration (Ctrough) of Glasdegib
Description: Ctrough of Glasdegib was measured in ng/mL.
Time Frame: Pre-dose: Cycle 1 Day 15 and Cycle 2 Day 1
Population: as for outcome 41
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | Non-intensive Study: Glasdegib + Azacitidine
Number analyzed (Participants) | 53
ng/ml
  Cycle 1 Day 15: number analyzed (Participants) | 34
  Cycle 1 Day 15 | 565.44 (126)
  Cycle 2 Day 1: number analyzed (Participants) | 37
  Cycle 2 Day 1 | 472.42 (122)

43. Secondary Outcome: Intensive Study: Number of Participants With Shift From Baseline in Corrected QT (QTc) Interval
Description: Triplicate 12-lead ECG measurements (each recording separated by approximately 2 minutes) were performed and average was calculated. The time corresponding to beginning of depolarization to repolarization of the ventricles (QT interval) was adjusted for RR interval using QT and RR from each ECG by Fridericia's formula (QTcF = QT divided by cube root of RR) and by Bazette's formula (QTcB = QT divided by square root of RR). Participants with maximum increase from baseline of <=450 to >500 msec (post-baseline) were summarized. Number of participants with shift from baseline for QTc were assessed. Only those QTc parameters in which at least 1 participant had data were reported.
Time Frame: Day 1 up to maximum of 2 years
Population: SA set included all participants who received at least one dose of study drug. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "Number Analyzed" signifies participants evaluable for specific time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive Study: Glasdegib + Cytarabine + Daunorubicin | Intensive Study: Placebo + Cytarabine + Daunorubicin
Number analyzed (Participants) | 188 | 189
Participants
  QTcB: <=450 msec (baseline) to <=450 msec (post-baseline): number analyzed (Participants) | 188 | 188
  QTcB: <=450 msec (baseline) to <=450 msec (post-baseline) | 51 | 71
  QTcB: <=450 msec (baseline) to >450-<=480 msec (post-baseline): number analyzed (Participants) | 188 | 188
  QTcB: <=450 msec (baseline) to >450-<=480 msec (post-baseline) | 64 | 63
  QTcB: <=450 msec (baseline) to >480-<=500 msec (post-baseline): number analyzed (Participants) | 188 | 188
  QTcB: <=450 msec (baseline) to >480-<=500 msec (post-baseline) | 18 | 11
  QTcB: <=450 msec (baseline) to >500 msec (post-baseline): number analyzed (Participants) | 188 | 188
  QTcB: <=450 msec (baseline) to >500 msec (post-baseline) | 11 | 6
  QTcB: >450-<=480 msec (baseline) to <=450 msec (post-baseline): number analyzed (Participants) | 188 | 188
  QTcB: >450-<=480 msec (baseline) to <=450 msec (post-baseline) | 2 | 3
  QTcB: >450-<=480 msec (baseline) to >450-<=480 msec (post-baseline): number analyzed (Participants) | 188 | 188
  QTcB: >450-<=480 msec (baseline) to >450-<=480 msec (post-baseline) | 20 | 17
  QTcB: >450-<=480 msec (baseline) to >480-<=500 msec (post-baseline): number analyzed (Participants) | 188 | 188
  QTcB: >450-<=480 msec (baseline) to >480-<=500 msec (post-baseline) | 16 | 10
  QTcB: >450-<=480 msec (baseline) to >500 msec (post-baseline): number analyzed (Participants) | 188 | 188
  QTcB: >450-<=480 msec (baseline) to >500 msec (post-baseline) | 1 | 5
  QTcB: >480-<=500 msec (baseline) to >450-<=480 msec (post-baseline): number analyzed (Participants) | 188 | 188
  QTcB: >480-<=500 msec (baseline) to >450-<=480 msec (post-baseline) | 1 | 0
  QTcB: >480-<=500 msec (baseline) to >480-<=500 msec (post-baseline): number analyzed (Participants) | 188 | 188
  QTcB: >480-<=500 msec (baseline) to >480-<=500 msec (post-baseline) | 2 | 1
  QTcB: >480-<=500 msec (baseline) to >500 msec (post-baseline): number analyzed (Participants) | 188 | 188
  QTcB: >480-<=500 msec (baseline) to >500 msec (post-baseline) | 1 | 0
  QTcB: >500 msec (baseline) to >500 msec (post-baseline): number analyzed (Participants) | 188 | 188
  QTcB: >500 msec (baseline) to >500 msec (post-baseline) | 1 | 1
  QTcF: <=450 msec (baseline) to <=450 msec (post-baseline): number analyzed (Participants) | 187 | 189
  QTcF: <=450 msec (baseline) to <=450 msec (post-baseline) | 116 | 132
  QTcF: <=450 msec (baseline) to >450-<=480 msec (post-baseline): number analyzed (Participants) | 187 | 189
  QTcF: <=450 msec (baseline) to >450-<=480 msec (post-baseline) | 50 | 39
  QTcF: <=450 msec (baseline) to >480-<=500 msec (post-baseline): number analyzed (Participants) | 187 | 189
  QTcF: <=450 msec (baseline) to >480-<=500 msec (post-baseline) | 8 | 10
  QTcF: <=450 msec (baseline) to >500 msec (post-baseline): number analyzed (Participants) | 187 | 189
  QTcF: <=450 msec (baseline) to >500 msec (post-baseline) | 5 | 0
  QTcF: >450-<=480 msec (baseline) to <=450 msec (post-baseline): number analyzed (Participants) | 187 | 189
  QTcF: >450-<=480 msec (baseline) to <=450 msec (post-baseline) | 2 | 1
  QTcF: >450-<=480 msec (baseline) to >450-<=480 msec (post-baseline): number analyzed (Participants) | 187 | 189
  QTcF: >450-<=480 msec (baseline) to >450-<=480 msec (post-baseline) | 5 | 5
  QTcF: >450-<=480 msec (baseline) to >500 msec (post-baseline): number analyzed (Participants) | 187 | 189
  QTcF: >450-<=480 msec (baseline) to >500 msec (post-baseline) | 1 | 1
  QTcF: >480-<=500 msec (baseline) to >480-<=500 msec (post-baseline): number analyzed (Participants) | 187 | 189
  QTcF: >480-<=500 msec (baseline) to >480-<=500 msec (post-baseline) | 0 | 1

44. Secondary Outcome: Non-intensive Study: Number of Participants With Shift From Baseline in Corrected QT (QTc) Interval
Description: as for outcome 43
Time Frame: Day 1 up to maximum of 3 years
Population: as for outcome 43
Measure: Count of Participants; unit: Participants
Arm/Group | Non-intensive Study: Glasdegib + Azacitidine | Non-intensive Study: Placebo + Azacitidine
Number analyzed (Participants) | 158 | 155
Participants
  QTcB: <=450 msec (baseline) to <=450 msec (post-baseline) | 48 | 58
  QTcB: <=450 msec (baseline) to >450-<=480 msec (post-baseline) | 53 | 43
  QTcB: <=450 msec (baseline) to >480-<=500 msec (post-baseline) | 6 | 11
  QTcB: <=450 msec (baseline) to >500 msec (post-baseline) | 7 | 3
  QTcB: >450-<=480 msec (baseline) to <=450 msec (post-baseline) | 0 | 1
  QTcB: >450-<=480 msec (baseline) to >450-<=480 msec (post-baseline) | 20 | 22
  QTcB: >450-<=480 msec (baseline) to >480-<=500 msec (post-baseline) | 13 | 8
  QTcB: >450-<=480 msec (baseline) to >500 msec (post-baseline) | 5 | 3
  QTcB: >480-<=500 msec (baseline) to >450-<=480 msec (post-baseline) | 1 | 2
  QTcB: >480-<=500 msec (baseline) to >480-<=500 msec (post-baseline) | 3 | 1
  QTcB: >480-<=500 msec (baseline) to >500 msec (post-baseline) | 2 | 3
  QTcF: <=450 msec (baseline) to <=450 msec (post-baseline): number analyzed (Participants) | 155 | 155
  QTcF: <=450 msec (baseline) to <=450 msec (post-baseline) | 100 | 104
  QTcF: <=450 msec (baseline) to >450-<=480 msec (post-baseline): number analyzed (Participants) | 155 | 155
  QTcF: <=450 msec (baseline) to >450-<=480 msec (post-baseline) | 39 | 36
  QTcF: <=450 msec (baseline) to >480-<=500 msec (post-baseline): number analyzed (Participants) | 155 | 155
  QTcF: <=450 msec (baseline) to >480-<=500 msec (post-baseline) | 7 | 0
  QTcF: >450 - <=480 (baseline) to <=450msec (post-baseline): number analyzed (Participants) | 155 | 155
  QTcF: >450 - <=480 (baseline) to <=450msec (post-baseline) | 1 | 1
  QTcF: >450 - <=480 msec (baseline) to >450 - <=480msec(post baseline) | 0 | 1
  QTcF: >450 - <=480 msec (baseline) to >480 - <=500 msec (post baseline) | 5 | 8
  QTcF: >480 msec (baseline) to <=500 msec (post baseline) | 1 | 4
  QTcF: >450 - <=480 (baseline) to >500 msec (post baseline) | 1 | 1
  QTcF: >480 - <=500msec (baseline) to >480 - <=500 msec (post baseline) | 1 | 0

ADVERSE EVENTS:
Time Frame: Intensive study: Day 1 up to maximum of 2 years; non-intensive study: Day 1 up to maximum of 3 years
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. All-Cause Mortality was assessed for all randomized participants whereas serious and other adverse events were assessed for safety population.
Arm/Group | Intensive Study: Glasdegib + Cytarabine + Daunorubicin | Intensive Study: Placebo + Cytarabine + Daunorubicin | Non-intensive Study: Glasdegib + Azacitidine | Non-intensive Study: Placebo + Azacitidine
All-Cause Mortality (participants affected / at risk) | 90/201 | 88/203 | 117/163 | 113/162
Serious Adverse Events (participants affected / at risk) | 86/198 | 92/201 | 117/162 | 124/160
Other Adverse Events (participants affected / at risk) | 194/198 | 195/201 | 154/162 | 148/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intensive Study: Glasdegib + Cytarabine + Daunorubicin (N=198) | Intensive Study: Placebo + Cytarabine + Daunorubicin (N=201) | Non-intensive Study: Glasdegib + Azacitidine (N=162) | Non-intensive Study: Placebo + Azacitidine (N=160)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 6 | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 18 | 17 | 24 | 20
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 3 | 2 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 1 | 1 | 2
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 2
Cardiac failure (Cardiac disorders) | 0 | 1 | 0 | 3
Cardiac failure acute (Cardiac disorders) | 1 | 0 | 1 | 0
Myocarditis (Cardiac disorders) | 1 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 4 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 3 | 2
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 0 | 2 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Neutropenic colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Disease progression (General disorders) | 2 | 5 | 14 | 22
Multiple organ dysfunction syndrome (General disorders) | 0 | 1 | 2 | 0
Pyrexia (General disorders) | 4 | 6 | 11 | 11
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 0 | 0 | 1
Arthritis infective (Infections and infestations) | 1 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 4 | 2 | 3 | 4
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 1 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 2 | 7
Clostridium difficile colitis (Infections and infestations) | 1 | 1 | 1 | 0
Enterobacter bacteraemia (Infections and infestations) | 0 | 1 | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 1 | 1 | 1
Infection (Infections and infestations) | 3 | 0 | 1 | 5
Neutropenic sepsis (Infections and infestations) | 1 | 2 | 3 | 5
Perirectal abscess (Infections and infestations) | 0 | 1 | 1 | 0
Pneumonia (Infections and infestations) | 15 | 11 | 29 | 36
Pneumonia fungal (Infections and infestations) | 2 | 2 | 2 | 0
Pseudomembranous colitis (Infections and infestations) | 1 | 0 | 0 | 1
Sepsis (Infections and infestations) | 15 | 13 | 14 | 10
Septic shock (Infections and infestations) | 2 | 4 | 4 | 7
Soft tissue infection (Infections and infestations) | 1 | 0 | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 9 | 4
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2
Blood creatinine increased (Investigations) | 3 | 1 | 2 | 2
Electrocardiogram QT prolonged (Investigations) | 13 | 8 | 5 | 3
Platelet count decreased (Investigations) | 1 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 3 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 2 | 2 | 1 | 1
Syncope (Nervous system disorders) | 1 | 0 | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 3 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 1
Hypotension (Vascular disorders) | 1 | 1 | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Splenic necrosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0
Intracardiac mass (Cardiac disorders) | 0 | 1 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Intussusception (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Graft versus host disease (Immune system disorders) | 0 | 1 | 0 | 0
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 1 | 0 | 0 | 0
Graft versus host disease in skin (Immune system disorders) | 1 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Anorectal infection (Infections and infestations) | 0 | 1 | 0 | 0
Atypical pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Brain abscess (Infections and infestations) | 0 | 1 | 0 | 0
Candida pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Clostridial sepsis (Infections and infestations) | 1 | 0 | 0 | 1
Clostridium bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Clostridium colitis (Infections and infestations) | 1 | 0 | 0 | 0
Device related bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 1 | 0 | 0
Disseminated varicella zoster virus infection (Infections and infestations) | 0 | 1 | 0 | 0
Enterococcal bacteraemia (Infections and infestations) | 2 | 0 | 1 | 1
Escherichia sepsis (Infections and infestations) | 1 | 1 | 0 | 0
Febrile infection (Infections and infestations) | 0 | 1 | 0 | 0
Fungal infection (Infections and infestations) | 1 | 0 | 0 | 0
Fungal sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Groin abscess (Infections and infestations) | 1 | 0 | 0 | 0
Herpes ophthalmic (Infections and infestations) | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 0 | 0
Pseudomonal bacteraemia (Infections and infestations) | 3 | 0 | 0 | 0
Pseudomonal sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0 | 0 | 0
Streptococcal sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Urethritis (Infections and infestations) | 1 | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 2 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 2 | 3 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 1
Adjustment disorder with depressed mood (Psychiatric disorders) | 1 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Embolism (Vascular disorders) | 0 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Mechanical ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Asthenia (General disorders) | 0 | 0 | 0 | 2
Death (General disorders) | 0 | 0 | 4 | 2
Sudden death (General disorders) | 0 | 0 | 1 | 1
Fatigue (General disorders) | 0 | 0 | 1 | 1
General physical health deterioration (General disorders) | 0 | 0 | 0 | 3
Soft tissue inflammation (General disorders) | 0 | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 1 | 0
Abscess (Infections and infestations) | 0 | 0 | 0 | 1
Anal abscess (Infections and infestations) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 2 | 4
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 2 | 4
Candida sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Catheter site infection (Infections and infestations) | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1
Herpes dermatitis (Infections and infestations) | 0 | 0 | 0 | 1
Infected skin ulcer (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 0 | 0 | 2
Liver abscess (Infections and infestations) | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Lower respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Otitis media acute (Infections and infestations) | 0 | 0 | 0 | 1
Periodontitis (Infections and infestations) | 0 | 0 | 0 | 2
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 0 | 0 | 0 | 1
Post procedural infection (Infections and infestations) | 0 | 0 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1 | 2
Rectal abscess (Infections and infestations) | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Subdiaphragmatic abscess (Infections and infestations) | 0 | 0 | 1 | 0
Suspected COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1
Systemic infection (Infections and infestations) | 0 | 0 | 0 | 1
Systemic mycosis (Infections and infestations) | 0 | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 2
Creatinine renal clearance decreased (Investigations) | 0 | 0 | 1 | 0
Electroencephalogram abnormal (Investigations) | 0 | 0 | 1 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Differentiation syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Central nervous system lesion (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 2 | 2
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 2 | 2
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 0 | 0 | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Partial seizures (Nervous system disorders) | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 2 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Aneurysm ruptured (Vascular disorders) | 0 | 0 | 0 | 1
Axillary vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 0 | 1 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 1 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiorenal syndrome (Cardiac disorders) | 0 | 0 | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Glossitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oral infection (Infections and infestations) | 0 | 0 | 1 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 1 | 0
Superficial vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Enteritis infectious (Infections and infestations) | 0 | 0 | 0 | 1
Epididymitis (Infections and infestations) | 0 | 0 | 0 | 1
Superinfection bacterial (Infections and infestations) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intensive Study: Glasdegib + Cytarabine + Daunorubicin (N=198) | Intensive Study: Placebo + Cytarabine + Daunorubicin (N=201) | Non-intensive Study: Glasdegib + Azacitidine (N=162) | Non-intensive Study: Placebo + Azacitidine (N=160)
Anaemia (Blood and lymphatic system disorders) | 101 | 97 | 73 | 71
Febrile neutropenia (Blood and lymphatic system disorders) | 97 | 96 | 23 | 22
Leukopenia (Blood and lymphatic system disorders) | 10 | 13 | 13 | 4
Neutropenia (Blood and lymphatic system disorders) | 41 | 43 | 38 | 30
Thrombocytopenia (Blood and lymphatic system disorders) | 52 | 52 | 38 | 35
Abdominal pain (Gastrointestinal disorders) | 31 | 29 | 12 | 10
Constipation (Gastrointestinal disorders) | 71 | 61 | 58 | 52
Diarrhoea (Gastrointestinal disorders) | 96 | 88 | 39 | 32
Haemorrhoids (Gastrointestinal disorders) | 13 | 19 | 9 | 11
Nausea (Gastrointestinal disorders) | 110 | 106 | 58 | 44
Vomiting (Gastrointestinal disorders) | 57 | 40 | 35 | 32
Asthenia (General disorders) | 15 | 11 | 16 | 18
Fatigue (General disorders) | 31 | 32 | 14 | 23
Oedema peripheral (General disorders) | 25 | 32 | 11 | 19
Pyrexia (General disorders) | 84 | 84 | 42 | 38
Pneumonia (Infections and infestations) | 32 | 33 | 19 | 16
Upper respiratory tract infection (Infections and infestations) | 9 | 11 | 12 | 11
Urinary tract infection (Infections and infestations) | 5 | 11 | 17 | 10
Alanine aminotransferase increased (Investigations) | 39 | 53 | 14 | 12
Aspartate aminotransferase increased (Investigations) | 30 | 41 | 11 | 9
Blood creatinine increased (Investigations) | 18 | 13 | 20 | 13
Electrocardiogram QT prolonged (Investigations) | 21 | 20 | 20 | 19
Gamma-glutamyltransferase increased (Investigations) | 12 | 22 | 10 | 8
Neutrophil count decreased (Investigations) | 56 | 49 | 22 | 23
Platelet count decreased (Investigations) | 77 | 73 | 30 | 26
Weight decreased (Investigations) | 21 | 22 | 36 | 19
White blood cell count decreased (Investigations) | 63 | 53 | 17 | 18
Decreased appetite (Metabolism and nutrition disorders) | 52 | 41 | 45 | 21
Hyperglycaemia (Metabolism and nutrition disorders) | 10 | 10 | 6 | 9
Hypoalbuminaemia (Metabolism and nutrition disorders) | 32 | 30 | 11 | 13
Hypocalcaemia (Metabolism and nutrition disorders) | 25 | 17 | 10 | 13
Hypokalaemia (Metabolism and nutrition disorders) | 76 | 83 | 35 | 22
Hypomagnesaemia (Metabolism and nutrition disorders) | 29 | 24 | 11 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 24 | 15 | 17 | 9
Hypophosphataemia (Metabolism and nutrition disorders) | 42 | 44 | 10 | 15
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 14 | 11 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 22 | 17 | 8 | 12
Muscle spasms (Musculoskeletal and connective tissue disorders) | 20 | 3 | 31 | 4
Dizziness (Nervous system disorders) | 23 | 18 | 9 | 14
Dysgeusia (Nervous system disorders) | 39 | 20 | 38 | 8
Headache (Nervous system disorders) | 39 | 47 | 4 | 9
Insomnia (Psychiatric disorders) | 27 | 30 | 12 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 23 | 23 | 10 | 20
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 | 23 | 12 | 18
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 19 | 20 | 8 | 11
Alopecia (Skin and subcutaneous tissue disorders) | 22 | 26 | 20 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 12 | 11 | 8 | 9
Rash (Skin and subcutaneous tissue disorders) | 46 | 51 | 10 | 13
Sinus tachycardia (Cardiac disorders) | 11 | 7 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 12 | 9 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 12 | 5 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 14 | 6 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 29 | 41 | 0 | 0
Chills (General disorders) | 20 | 11 | 0 | 0
Mucosal inflammation (General disorders) | 12 | 7 | 0 | 0
Non-cardiac chest pain (General disorders) | 13 | 8 | 0 | 0
Oedema (General disorders) | 9 | 19 | 0 | 0
Bacteraemia (Infections and infestations) | 16 | 11 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 14 | 13 | 0 | 0
Blood bilirubin increased (Investigations) | 25 | 13 | 0 | 0
Lymphocyte count decreased (Investigations) | 19 | 21 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 13 | 9 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 15 | 11 | 0 | 0
Paraesthesia (Nervous system disorders) | 11 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 19 | 19 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 13 | 10 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 8 | 11 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 21 | 21 | 0 | 0
Hypertension (Vascular disorders) | 10 | 25 | 0 | 0
Hypotension (Vascular disorders) | 18 | 17 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 12 | 7
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 11 | 1
C-reactive protein increased (Investigations) | 0 | 0 | 7 | 9
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 11 | 10
White blood cell count increased (Investigations) | 0 | 0 | 9 | 8
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 9 | 5

LIMITATIONS AND CAVEATS:
In this study, inadvertently a participant was counted twice for an non-SAE "Pyrexia" at PCD, at SCD update this duplicity has been rectified. Due to this reason total number of participants affected by non-SAE in non-intensive placebo arm was updated to "148".

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-04-12): https://cdn.clinicaltrials.gov/large-docs/79/NCT03416179/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-14): https://cdn.clinicaltrials.gov/large-docs/79/NCT03416179/SAP_001.pdf